#### The GlaxoSmithKline group of companies

| Division | : ' | Worldwide Development |
|-------------------------|-----|-----------------------------------|
| <b>Information Type</b> | : ] | Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for 204716
A 24-week, Phase III, open-label, non-comparative, multicenter study to evaluate efficacy and safety of GSK1278863 in Japanese hemodialysis subjects with anemia associated with chronic kidney disease who are not taking erythropoiesis stimulating agents.

Compound Number : GSK1278863

Effective Date : 29-Nov-2017

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 204716.
- This RAP is intended to describe the 204716 analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| PPD | 29-Nov-2017 |
|-------------------------------------------------------|--------------|
| Biostatistics Group 2, Biomedical Data Sciences Japan | 29-1NOV-2017 |

#### Approved by:

| PPD | | 29-Nov-2017 |
|---|---|---|
| Manager, Biostatistics Group 2, Biomedical Data Sciences Japan | | 29-110V-2017 |
| PPD | | |
| Manager, Sta | tistical Programming & Reporting Group, Biomedical | 29-Nov-2017 |
| Data Sciences Japan | | |

#### **Revision History (Appendix 16):**

| Version | Date |
|---------------------------------------------------------|-------------|
| Reporting and Analysis Plan_204716_Final_V1.0 | 19-Jun-2017 |
| Reporting and Analysis Plan_204716_Amendment_Final_V1.1 | 11-Oct-2017 |
| Reporting and Analysis Plan_204716_Amendment_Final_V1.2 | 29-Nov-2017 |


### The GlaxoSmithKline group of companies

204716

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorized copying or use of this information is prohibited.

#### **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | REPC | ORTING & ANALYSIS PLAN SYNOPSIS | 6 |
| 2. | SUMN<br>2.1.<br>2.2.<br>2.3.<br>2.4. | MARY OF KEY PROTOCOL INFORMATION Changes to the Protocol Defined Statistical Analysis Plan Study Objective(s) and Endpoint(s) Study Design Statistical Hypotheses | 8<br>8<br>10 |
| 3. | PLAN<br>3.1.<br>3.2. | NED ANALYSESInterim AnalysesFinal Analyses | 11 |
| 4. | ANAL<br>4.1. | YSIS POPULATIONSProtocol Deviations | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING<br>/ENTIONS | 13 |
| 6. | STUD<br>6.1. | Y POPULATION ANALYSES Overview of Planned Analyses | 14 |
| 7. | PRIMA | ARY STATISTICAL ANALYSES Primary Efficacy Analyses 7.1.1. Overview of Planned Primary Efficacy Analyses 7.1.2. Planned Efficacy Statistical Analyses 7.1.3. Planned Summary Display Details | 19<br>19<br>19 |
| 8. | SECC<br>8.1. | ONDARY STATISTICAL ANALYSES | 22<br>22<br>24 |
| | 8.2. | Safety Analyses | 29<br>29<br>32 |
| | 8.3. | Pharmacokinetic Analyses 8.3.1. Overview of Planned Pharmacokinetic Analyses 8.3.2. Drug Concentration Measures 8.3.3. Pharmacokinetic Parameters 8.3.4. Population Pharmacokinetic (PopPK) Analyses | 36<br>36<br>36 |
| | 8.4.<br>8.5. | Pharmacokinetic / Pharmacodynamic Analyses Pharmacokinetic / Pharmacodynamic Analyses | 38 |
| 9. | REFE | RENCES | 39 |


| ١0. | APPE | NDICES | 40 |
|---|---|---|---|
| | 10.1. | Appendix 1: Protocol Deviation Management and Definitions for Per | |
| | | Protocol Population | 41 |
| | 10.2. | Appendix 2: Time & Events | 42 |
| | | 10.2.1. Protocol Defined Time & Events | 42 |
| | 10.3. | Appendix 3: Assessment Windows | 44 |
| | | 10.3.1. Definitions of Analysis Time Point | 44 |
| | 10.4. | Appendix 4: Treatment States and Phases | |
| | | 10.4.1. Treatment States | |
| | 10.5. | Appendix 5: Data Display Standards & Handling Conventions | 47 |
| | | 10.5.1. Study Treatment & Sub-group Display Descriptors | |
| | | 10.5.2. Baseline Definition & Derivations | |
| | | 10.5.3. Reporting Process & Standards | |
| | 10.6. | Appendix 6: Derived and Transformed Data | |
| | | 10.6.1. General | |
| | | 10.6.2. Study Population | |
| | | 10.6.3. Efficacy | |
| | | 10.6.4. Safety | |
| | | 10.6.5. Pharmacokinetic | |
| | 10.7. | Appendix 7: Premature Withdrawals & Handling of Missing Data | |
| | | 10.7.1. Premature Withdrawals | |
| | | 10.7.2. Handling of Missing Data | 60 |
| | 10.8. | Appendix 8: Values of Potential Clinical Importance | 61 |
| | | 10.8.1. Laboratory Values | |
| | | 10.8.2. Vital Signs | |
| | 10.9. | Appendix 9: Multicenter Studies | |
| | 10.10. | Appendix 10: Examination of Covariates, Subgroups & Other Strata | |
| | | 10.10.1. Handling of Covariates, Subgroups & Other Strata | |
| | 10.11. | Appendix 11: Multiple Comparisons & Multiplicity | |
| | | 10.11.1. Handling of Multiple Comparisons & Multiplicity | 64 |
| | 10.12. | Appendix 12: Model Checking and Diagnostics for Statistical | |
| | | Analyses | |
| | 10.13. | Appendix 13 – Abbreviations & Trade Marks | |
| | | 10.13.1. Abbreviations | |
| | | 10.13.2. Trademarks | |
| | 10.14. | Appendix 14: List of Data Displays | |
| | | 10.14.1. Data Display Numbering | |
| | | 10.14.2. Mock Example Shell Referencing | |
| | | 10.14.3. Study Population Tables | |
| | | 10.14.4. Efficacy Tables | |
| | | 10.14.5. Efficacy Figures | |
| | | 10.14.6. Safety Tables | |
| | | 10.14.7. Safety Figures | |
| | | 10.14.8. Pharmacokinetic Tables | |
| | | 10.14.9. Pharmacokinetic Figures | |
| | | 10.14.10.ICH Listings | |
| | | 10.14.11. Non-ICH Listings | |
| | 10 15 | 10.14.12. Patient Profile Listings | |
| | | Appendix 15: Example Mock Shells for Data Displays | |
| | 10.10. | Appendix 16: RAP Amendment(s) | 99 |


### 1. REPORTING & ANALYSIS PLAN SYNOPSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | <ul> <li>This RAP describes the planned analyses and outputs required for the final<br/>Clinical Study Report (CSR) for study 204716.</li> </ul> |
| Protocol | Protocol This RAP is based on the protocol amendment v04 (Dated: 19/Jul/2017) of study 204716 (GSK Document No.2015N266250_04]. |
| Primary<br>Objective | To characterize the appropriateness of the starting dose of GSK1278863 in HD patients not using ESAs |
| Primary | Change from baseline in Hgb at Week 4 |
| Endpoint | <ul> <li>Number (%) of subjects by Hgb change from baseline category at Week 4</li> </ul> |
| Study<br>Design | This is a 24-week, Phase III, open-label, non-comparative, multi-center study to evaluate efficacy and safety of GSK1278863 in approximately 22 Japanese hemodialysis subjects with anemia associated with chronic kidney disease who are not taking erythropoiesis stimulating agents. |
| Planned | No interim analysis is planned. |
| Analyses | <ul> <li>Final analyses will be performed according to the steps described in Section<br/>3.2.</li> </ul> |
| | <ul> <li>All decisions regarding final analyses, as defined in this RAP document, will be<br/>made prior to Database Freeze of the study data.</li> </ul> |
| Analysis<br>Populations | All Screening Population will consist of all subjects who are given subject number and are collected data at screening. |
| | <ul> <li>Enrolled Population will consist of subjects in 'All Screening' except for screen<br/>failures (who never passed screening even if rescreened).</li> </ul> |
| | <ul> <li>Assigned Population will consist of all randomized subjects regardless of study<br/>treatment actually received or not</li> </ul> |
| | <ul> <li>All Treated Subjects Population will consist of all subjects who receive at least<br/>one dose of GSK1278863.</li> </ul> |
| | <ul> <li>Pharmacokinetic (PK) Population will consist of all subjects who received<br/>GSK1278863 with the PK samples collected and analysed.</li> </ul> |
| Hypothesis | This single arm study is a study with an aim of an estimation. The primary objective of this study is to evaluate the initial anemia correction of GSK1278863 in HD patients not using ESAs. There will be no hypothesis testing performed in this study. |
| Primary Analyses For the change from baseline in Hgb at Week 4, the summary statis calculated, along with the two-sided 95% confidence interval based distribution. | |
| | • The change in Hgb at Week 4 will be classified into different categories (i.e., ≤- |


| Overview | Key Elements of the RAP |
|---|---|
| | 2, >-2 to -1, >-1 to 0, >0 to 1, >1 to 2, and >2 g/dL), and the number (%) of |
| | subjects in each category will be summarized. |

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

### 2.1. Changes to the Protocol Defined Statistical Analysis Plan

No changes from the originally planned statistical analysis specified in the protocol amendment v04 (Dated: 19/Jul/2017) are present.

### 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary | , |
| To characterize the appropriateness of<br>the starting dose of GSK1278863 in HD<br>patients not using ESAs Secondary | <ul> <li>Change from baseline in Hgb at Week 4</li> <li>Number (%) of subjects by Hgb change from baseline category at Week 4</li> </ul> |
| To characterize overall Hgb control of<br>GSK1278863 in HD patients not using<br>ESAs | <ul> <li>Hgb and changes from baseline</li> <li>Number (%) of subjects who have a Hgb level within the target range (10.0–12.0 g/dL)</li> <li>Time (in days) to reach the lower target Hgb level (10.0 g/dL)</li> <li>Number (%) of subjects who have a Hgb level of less than &lt; 7.5 g/dL</li> <li>Number (%) of subjects who have a Hgb increase of more than &gt; 2-g/dL over any 4 weeks</li> <li>Number (%) of subjects who have a Hgb level of more than &gt; 13.0 g/dL and number of episodes</li> </ul> |
| To characterize the pharmacokinetics of<br>GSK1278863 | AUC and Cmax of plasma GSK1278863 |
| <ul> <li>To characterize the effect on iron use of<br/>GSK1278863 in HD patients not using<br/>ESAs</li> <li>To characterize the effect on iron<br/>metabolism of GSK1278863 in HD<br/>patients not using ESAs</li> </ul> | <ul> <li>Dose of intravenous iron</li> <li>Number (%) of subjects who used intravenous iron</li> <li>Change from baseline in ferritin</li> <li>Change from baseline in transferrin saturation</li> </ul> |

| Objectives | Endpoints |
|---|---|
| | Changes from baseline in hepcidin, serum iron, and total iron binding capacity (TIBC) |
| To characterize dose adjustment of<br>GSK1278863 in HD patients not using<br>ESAs | <ul> <li>Distribution of dose level</li> <li>Frequency of dose adjustments</li> <li>Duration of treatment interruption due to Hgb &gt; 13 g/dL</li> </ul> |
| Safety | |
| To assess the safety and tolerability of<br>GSK1278863 in HD patients not using<br>ESAs | <ul> <li>Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), including adverse events of special interest (AESIs)</li> <li>Reasons for discontinuation of study medication</li> <li>Laboratory tests, electrocardiogram (ECG), vital signs, and ophthalmology assessments</li> </ul> |

#### 2.3. Study Design



#### 2.4. Statistical Hypotheses

This single arm study is a study with an aim of an estimation. The primary objective of this study is to evaluate the initial anemia correction of GSK1278863 in HD patients not

using ESAs. There will be no hypothesis testing performed in this study. Two-sided 95% confidence intervals will be used for efficacy estimation.

#### 3. PLANNED ANALYSES

#### 3.1. Interim Analyses

No interim analysis is planned.

#### 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. All criteria for releasing the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Population Definition / Criteria | |
|---|---|---|
| All Screening | <ul> <li>Consists of all subjects who are given subject<br/>number and are corrected data at screening.</li> </ul> | Study Population |
| Enrolled | Consist of subjects in 'All Screening' except for<br>screen failure (who never passed screening<br>even if rescreened). | <ul> <li>Study Population<br/>(some displays for<br/>EudraCT)</li> </ul> |
| Assigned | Consist of all subjects who are given<br>randomization number regardless of whether<br>they actually receive GSK1278863. | Study Population |
| All Treated<br>Subjects | Consist of all subjects who received at least one dose of GSK1278863. | <ul><li>Study Population</li><li>Efficacy</li><li>Safety</li></ul> |
| PK | Consist of all subjects who received<br>GSK1278863 with the PK samples collected<br>and analyzed. | • PK |

#### NOTES:

- Basically, enrolled population will be the same as assigned population because a subject is going to be given randomized number as soon as passed screening
- Please refer to Appendix 14: List of Data Displays which details the population to be used for each displays being generated.

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorized on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 10.2 | Appendix 2: Time & Events |
| 10.3 | Appendix 3: Assessment Windows |
| 10.4 | Appendix 4: Treatment States and Phases |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.6 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| 10.8 | Appendix 8: Values of Potential Clinical Importance |
| 10.9 | Appendix 9: Multicenter Studies |
| 10.10 | Appendix 10: Examination of Covariates, Subgroups & Other Strata |
| 10.11 | Appendix 11: Multiple Comparisons & Multiplicity |
| 10.12 | Appendix 12: Model Checking and Diagnostics for Statistical Analyses. |

#### 6. STUDY POPULATION ANALYSES

#### 6.1. Overview of Planned Analyses

The study population analyses will be based on the All Treated Subjects population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Endpoint / Parameter / Display Type | Population | Data D | isplays G | enerated |
|---|---|---|---|---|
| | | Table | Figure | Listing |
| Subject Disposition | | | | |
| Subject Status and Reason for Study Withdrawal | Assigned | Υ | | |
| Subject Status and Reason for Study Withdrawal by Dialysis Status | Assigned | Y | | |
| Reasons for Subject Withdrawal | Assigned | | | Υ |
| Treatment Status and Reasons for Discontinuation of Study Treatment | All Treated | Y | | Υ |
| Screening Status and Reasons for Screen Failure | All Screening | Y | | Y |
| Subjects Enrolled by Country and Site ID | Enrolled | Y | | |
| Protocol Deviations | | | | |
| Important Protocol Deviations | Assigned | Υ | | Υ |
| Subjects with Inclusion/Exclusion Criteria Deviations | Assigned | Y | | Y |
| Populations Analyzed | | - | | |
| Study Populations | All Screening | Υ | | |
| Exclusions from Study Population | Assigned | Υ | | |
| Subjects Excluded from Any Population | Assigned | | | Y |
| <b>Demographic and Baseline Characteristics</b> | | | | |
| Demographic Characteristics | All Treated | Y | | Υ |
| Demographic Characteristics<br>by Dialysis Status | All Treated | Y | | |
| Age Ranges | Enrolled | Y | | |
| Race and Racial Combinations | All Treated | Υ | | Y [1] |
| Family History for CV Risk Factors | All Treated | Υ | | Y |
| Substance Use (History of Tobacco Use, Alcohol Intake) | All Treated | Υ | | Y |
| Prior and Concomitant Medications | | • | | |
| Current/Past Medical Conditions | All Treated | Υ | | Y |
| Current/Past Medical Conditions<br>by Dialysis Status | All Treated | Υ | | |
| Concomitant Medications [2] | All Treated | Y | | Y |
| Other Concomitant Medications [3] | All Treated | Y | | Y |

| Endpoint / Parameter / Display Type | Population | Data Displays Generated | | |
|---|---|---|---|---|
| | | Table | Figure | Listing |
| Other Concomitant Medications [3] by Dialysis Status | All Treated | Υ | | |
| Blood products and blood supportive care products [4] | All Treated | Υ | | Υ |
| Blood products and blood supportive care products [4] by Dialysis Status | All Treated | Υ | | |
| Dialysis | | | | |
| Dialysis Status | All Treated | Y | | Υ |
| Baseline Mode of Dialysis | All Treated | Υ | | Υ |
| Subjects with Change in Hemodialysis | All Treated | | | Υ |
| Baseline Vascular Access | All Treated | Υ | | Υ |
| Subjects with Vascular Therapeutic Procedures during the study period | All Treated | | | Y |
| Exposure and Treatment Compliance | | | | |
| Exposure to Study Treatment | All Treated | Υ | | Υ |
| Exposure to Study Treatment by Dialysis Status | All Treated | Y | | |
| Treatment Compliance | All Treated | Y | | Υ |

#### NOTES:

- Y = Yes display generated.
- Some summaries will be generated as efficacy analyses.
- [1] Listing of race.
- [2] Concomitant medications in prior-therapy period, on-therapy period, and post-therapy period will be summarized separately.
- [3] On-therapy ESA and iron medication will be provided.
- [4] On-therapy blood products and blood supportive care products will be provided.

#### 6.1.1. Planned Summary Display Details

A subject who has multiple subject numbers (i.e. rescreened subject) will be analyzed as a unique subject based on the latest screening result.

The definition of subgroup is described in Appendix 10.

#### • Subject Disposition

#### Subject Status and Reason for Study Withdrawal

The number and percentage of subjects completing the study or withdrawing early from the study will be summarized overall and by reason for withdrawal. Reasons for withdrawal will be listed for subject. The subgroup analysis for dialysis status will be summarized as the same.

Treatment Status and Reasons for Discontinuation of Study Treatment

The number and percentage of subjects completing the treatment or discontinuing the treatment during the study will be summarized overall and by reason.

#### Screening Status and Reasons for Screen Failure

The number and percentage of subjects who failed screening and were therefore not randomized into the study, overall and by reason, will be summarized for all screening population. Note that the reasons for rescreen subjects who initially failed but subsequently enrolled are not included in the display (see Section 10.6.2).

#### Subjects Enrolled by Country and Site ID

The number and percentage of subjects by region, country and center will be summarized

#### • Protocol Deviations

#### **Important Protocol Deviations**

The number and percentage of subjects who had important protocol deviations defined in PDMP will be summarized.

#### Subjects with Inclusion/Exclusion Criteria Deviations

The number and percentage of subjects with any Inclusion/Exclusion Criteria Deviations will be summarized, further classifying inclusion/exclusion deviations.

#### Population Analyzed

#### Study Populations

The number of subjects in each analysis population (defined in Section 4) will be summarized.

#### Exclusions from Study Population

The number of subjects excluded from All Treated Subjects population will be summarized for the assigned population.

#### • Demographic and Baseline Characteristics

#### Demographic Characteristics

The number and percentage of subjects or summary statistics will be provided for the demographic and baseline characteristics: Sex, Age (years), Age Group (years), Ethnicity, Race detail, Height, Weight, and Body Mass Index. Age Group (years) will be categorized into 3 ('<=18', '19-64', '>=65'). The subgroup analysis for dialysis status will be summarized as the same.

#### Age Ranges

The number and percentage of subjects within each age range category will be provided. Age range will be categorized into: Adult (18-64 years), >=65-84 years, >=85 years.

#### Race and Racial Combinations

Summaries of race and racial combinations will be provided.

#### Family History for CV Risk Factors

A summary of family (first degree relatives) history for CV risk factors will be provided.

#### Substance Use (History of Tobacco Use, Alcohol Intake)

A summary of substance use will be provided.

#### • Prior and Concomitant Medications

#### Current/Past Medical Conditions

The number and percentage of subjects with current and past medical conditions recorded in eCRF will be provided. The subgroup analysis for dialysis status will be summarized as the same.

#### Concomitant Medications

The number and percentage of subjects reporting the use of each concomitant medication will be summarized by anatomical therapeutic chemical (ATC) Level 1, and Ingredient. Summaries of pre-therapy, on-therapy, and post-therapy medication will be provided separately. See Section 10.4.1.3 for treatment states for concomitant medications.

#### Other concomitant medications

The similar summary as above will be provided focusing on on-therapy ESA and iron medication. See Section 10.4.1.3 for treatment states. The subgroup analysis for dialysis status will be summarized as the same.

#### Blood products and blood supportive care products

The number and percentage of subjects who use blood products and/or blood supportive care products will be provided. The details for the use will also be provided. The subgroup analysis for dialysis status will be summarized as the same.

#### Dialysis

#### Dialysis Status

The number and percentage of subjects with dialysis status of newly started dialysis and maintenance dialysis will be provided. Definitions of dialysis status are described in the protocol section 5.3.

#### Baseline Mode of Dialysis

The number and percentage of subjects with each baseline mode of dialysis (i.e. haemodialysis, haemofiltration, or haemodiafiltration) will be provided.

#### Baseline Vascular Access

The number and percentage of subjects with each baseline vascular access will be provided. Previous vascular access will be summarized as the same.

#### • Exposure and Treatment Compliance

#### Exposure to Study Treatment

Full details of exposure definition are presented in Appendix 6.

Daily dose, cumulative dose, and days on study drug will be summarized using mean, standard deviation, median, minimum, and maximum. Regarding days on study drug, the number and percentage of subjects within each category (i.e. 1-28, 29-56, 57-84, 85-112, 113-140, 141-168, >168 (days)) will also be provided. The subgroup analysis for dialysis status will be summarized as the same.

#### Treatment Compliance

Full details of treatment compliance definition are presented in Appendix 6.

The number and percentage of subjects within each category of treatment compliance will be provided and the categories will be classified into <80%, 80% to 120%, and >120%.

#### 7. PRIMARY STATISTICAL ANALYSES

#### 7.1. Primary Efficacy Analyses

#### 7.1.1. Overview of Planned Primary Efficacy Analyses

The primary efficacy analyses will be based on the All Treated Subjects population, unless otherwise specified.

Table 3 provides an overview of the planned efficacy analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 3 Overview of Planned Primary Efficacy Analyses

| Endpoint / Parameter/ Display Type | Absolute | | | | | | |
|---|---|---|---|---|---|---|---|
| | Sta | ts Anal | ysis | Sum | mary | Indiv | idual |
| | T | F | L | T | F | F | L |
| Change from baseline in Hgb at Week 4 | | | | Υ | | | |
| Number (%) of subjects by Hgb change from baseline | | | | Υ | | | |
| category at Week 4 [1] | | | | | | | |
| Change from baseline in Hgb at Week 4 | | | | Υ | | | |
| by Dialysis Status | | | | | | | |
| Number (%) of subjects by Hgb change from baseline | | | | Υ | | | |
| category at Week 4 [1] | | | | | | | |
| by Dialysis Status | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

 $[1] \le -2$ , -2 to -1, -1 to 0, 0 to 1, 1 to 2, and >2 g/dL. In addition, within  $\pm 1$  g/dL and over  $\pm 2$  g/dL.

#### 7.1.2. Planned Efficacy Statistical Analyses

#### **Primary Analyses**

#### Endpoint(s)

- Change from baseline in Hgb at Week 4
- Number (%) of subjects by Hgb change from baseline category at Week 4

#### **Model Specification**

- Hgb values from central laboratory will be used, unless otherwise specified. However, if a
  central laboratory Hgb value is missing, a corresponding non-missing HemoCue Hgb value will
  be used (See Section 10.6.3).
- The primary analysis is to assess modest increase in Hgb in initial response to GSK1278863
  (i.e., Hgb increase by ≤ 2 g/dL after 4 weeks of treatment), on the basis of the mean change
  from baseline in Hgb at Week 4 as well as the number (%) of subjects by Hgb change from
  baseline category at Week 4 as the primary efficacy endpoints.
- For the change from baseline in Hgb at Week 4, the summary statistics will be calculated,


204716

along with the two-sided 95% confidence interval based on t-distribution.

• The change in Hgb at Week 4 will be classifieds into different categories (i.e.,  $\leq$ -2, >-2 to - 1, >-1 to 0, >0 to 1, >1 to 2, and >2 g/dL), and the number (%) of subjects in each category will be summarized. In addition, 'within  $\pm$  1 g/dL (i.e.,  $\geq$ -1 and  $\leq$ 1 g/dL)' and 'over  $\pm$  2 g/dL (i.e., <-2 and >2 g/dL)' categories will be provided.

#### 7.1.3. Planned Summary Display Details

The definition of subgroup is described in Appendix 10.

#### Change from baseline in Hgb at Week 4

This summary will be included within a summary of change from baseline in Hgb at each assessment visit (See Section 8.1.2). The values will be summarized using mean, standard deviation, 95%CI, minimum, P25, median, P75, and maximum at Week 4 visit. The subgroup analysis will be summarized as the same.

#### Number (%) of subjects by Hgb change from baseline category at Week 4

The number and percentage of subjects within each category will be provided and the categories will be classified into  $\leq$ -2, >-2 to -1, >-1 to 0, >0 to 1, >1 to 2, and >2 g/dL). In addition, 'within  $\pm$  1 g/dL (i.e.,  $\geq$ -1 and  $\leq$ 1)' and 'over  $\pm$  2 g/dL (i.e., <-2 and >2)' categories will be provided. The subgroup analysis will be summarized as the same.

#### 8. SECONDARY STATISTICAL ANALYSES

#### 8.1. Secondary Efficacy Analyses

#### 8.1.1. Overview of Planned Secondary Efficacy Analyses

The secondary efficacy analyses will be based on the All Treated Subjects population, unless otherwise specified.

Table 4 provides an overview of the planned secondary efficacy analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 4 Overview of Planned Efficacy Analyses

| Endpoint / Parameter/ Display Type | Absolute | | | | | |
|---|---|---|---|---|---|---|
| , | Stats A | Analysis | Sum | mary | Indiv | /idual |
| | Т | F | Т | F | F | L |
| Hgb | • | | | | • | |
| Hgb at each assessment visit | | | Υ | Υ | | Υ |
| Hgb at each assessment visit | | | Υ | Υ | | |
| by Dialysis Status | | | | | | |
| Change from baseline at each assessment visit | | | Υ | Υ | | Υ |
| Change from baseline at each assessment visit | | | Υ | Υ | | |
| by Dialysis Status | | | | | | |
| Number (%) of subjects with Hgb within the target range | | | Υ | Υ | | |
| at each assessment visit [1] | | | | | | |
| Number (%) of subjects with Hgb within the target range | | | Υ | Υ | | |
| at each assessment visit [1] | | | | | | |
| by Dialysis Status | | | | | | |
| Time (in days) to reach the lower target Hgb level | Υ | Υ | | | | |
| (10.0 g/dL) [2] [3] | | | | | | |
| Time (in days) to reach the lower target Hgb level | Υ | Υ | | | | |
| (10.0 g/dL) [2] [3] | | | | | | |
| by Dialysis Status | | | | | | |
| Number (%) of subjects who have an Hgb level of less | | | Υ | | | Υ |
| than 7.5 g/dL [3] | | | | | | |
| Number (%) of subjects who have an Hgb level of less | | | Υ | | | |
| than 7.5 g/dL [3] | | | | | | |
| by Dialysis Status | | | | | | |
| Number (%) of subjects who have an Hgb increase of | | | Υ | | | Υ |
| more than 2.0 g/dL over any 4 weeks [3] | | | | | | |
| Number (%) of subjects who have an Hgb increase of | | | Υ | | | |
| more than 2.0 g/dL over any 4 weeks [3] | | | | | | |
| by Dialysis Status | | | | | | |
| Number (%) of subjects who have an Hgb level of more | | | Υ | | | Υ |
| than 13.0 g/dL and number of episodes [3] | | 1 | V | - | | |
| Number (%) of subjects who have an Hgb level of more | | | Υ | | | |
| than 13.0 g/dL and number of episodes [3] | | | | | | |
| by Dialysis Status | | - | | | | V |
| Hemocue Hgb | | | | | | Υ |

| Endpoint / Parameter/ Display Type | | | | | | |
|---|---|---|---|---|---|---|
| , | Stats A | nalysis | | olute<br>mary | Indiv | vidual |
| | T | F | T | T F | F | 1 |
| Scatter plot of Hgb assessments: Central Laboratory vs. HemoCue | | Y | | | | |
| | | | | <u> </u> | | |
| Iron use | | 1 | V | T | | T V |
| Dose of i.v. iron during the treatment period | <del> </del> | | Y | | | Y |
| Dose of i.v. iron during the treatment period by Dialysis Status | | | | | | |
| Number (%) of subjects who use iron during the treatment period | | | Υ | | | |
| Number (%) of subjects who use iron during the treatment period | | | Υ | | | |
| by Dialysis Status | | | | | | |
| Iron Parameters (ferritin, TSAT [4], hepcidin [4], serum i | ron, and | TIBC) | | | | |
| Raw observed value at each assessment visit | | | Υ | | | Υ |
| Raw observed value at each assessment visit | | | Y | | | <u> </u> |
| by Dialysis Status | | | - | | | |
| Change from baseline at each assessment visit | | | Υ | Υ | | |
| Change from baseline at each assessment visit | | | Υ | | | |
| by Dialysis Status | | | | | | |
| Dose adjustment [5] | | | | ı | | 1 |
| Dose level (mg) at each assessment visit | | | Υ | Υ | | Υ |
| Dose level (mg) at each assessment visit | | | Y | Y | | |
| by Dialysis Status | | | | | | |
| Duration (days) of treatment interruption due to Hgb | | | Υ | | | |
| >13.0 g/dL [3] | | | | | | |
| Duration (days) of treatment interruption due to Hgb | | | Υ | | | |
| >13.0 g/dL [3] | | | | | | |
| by Dialysis Status | | | | | | |
| Dose adjustment | | | Υ | | | |
| Dose adjustment | | | Υ | | | |
| by Dialysis Status | | | | | | |
| Number (%) of subjects with each dose level at each | | | Υ | | | |
| assessment visit | | | | | | |
| Number (%) of subjects with each dose level at each | | | Υ | | | |
| assessment visit | | | | | | |
| by Dialysis Status | | | | | | |
| Number of dose adjustment to reach the lower Hgb target Hgb level (10.0 g/dL) | | | Υ | | | |
| Number of dose adjustment to reach the lower Hgb target | | | Υ | | | |
| Hgb level (10.0 g/dL) | | | | | | |
| by Dialysis Status | | | | | | |
| Other | | | | | | |
| Scatter plot of change from baseline in Hgb at Week 4 vs. | | | | Υ | | |
| candidate covariates [6] | <u> </u> | <u> </u> | | | | |
| Scatter plot of mean dose vs. candidate covariates [6] | | | | Υ | | |
| NOTES . | | | | | | |

<sup>[1]</sup> Not only within the target range, but also subjects with above and below target range will be assessed.
[2] Time to first reach the lower target Hgb level will be estimated by Kaplan-Meier method using P25, median and P75. Subjects who could not reach lower target will be regarded as censored.

| Endpoint / Parameter/ Display Type | Absolute | | | | |
|---|---|---|---|---|---|
| | Stats Analysis Summary Individua | | | idual | |
| | T F | Т | F | F | L |

- [3] On-therapy Hgb values observed in scheduled visits will be included. On-therapy Hgb values observed in unscheduled visits will be included if specified (see Section 8.1.2)
- [4] Based on literature review the distributions of TSAT and hepcidin are skewed and require a log-transformation.
- [5] Summaries for dose adjustment will be based on HemoCue Hgb values including those of unscheduled visits.
- [6] Figures will include the candidate covariates of body weight and baseline Hgb, and will be produced for overall and dialysis status groups.

#### 8.1.2. Planned Efficacy Table Displays

#### • Hgb

#### Hgb at each assessment visit

The values will be summarized using mean, standard deviation, 95%CI, minimum, P25, median, P75, and maximum at each assessment visit. Graphical summaries will be provided using mean and 95% CI over time. The subgroup analysis for dialysis status will be summarized as the same.

#### Change from baseline at each assessment visit

The values will be summarized using mean, standard deviation, 95%CI, minimum, P25, median, P75, and maximum at each assessment visit. Graphical summaries will be provided using mean and 95% CI over time. This will be also summarized by baseline dialysis status.

#### Number (%) of subjects with Hgb within the target range at each assessment visit

The number and percentage of subjects with Hgb within, above and below the target range at each assessment visit will be summarized. This will be also summarized by baseline dialysis status.

#### Time (in days) to reach the lower target Hgb level (10.0 g/dL)

The time (in days) will be summarized using P25, median, and P75 by Kaplan-Meier method. Kaplan-Meier plot of time to event will be provided using on-therapy Hgb values. Subjects who could not reach lower target will be regarded as censored. This will be also summarized by baseline dialysis status.

#### Number (%) of subjects who have an Hgb level of less than 7.5 g/dL

The number and percentage of subjects who have an Hgb level of less than 7.5 g/dL will be summarized. On-therapy Hgb values observed in both scheduled and unscheduled visits will be included in the summary. This will be also summarized by baseline dialysis status.

## Number (%) of subjects who have an Hgb increase of more than 2.0 g/dL over any 4 weeks

The number and percentage of subjects who have an Hgb increase of more than 2.0 g/dL over any 4 weeks will be summarized. On-therapy Hgb values will be used for the summary. This will be also summarized by baseline dialysis status. See Section 10.6.3 for detailed derivation.

# Number (%) of subjects who have an Hgb level of more than 13.0 g/dL and number of episodes

The number and percentage of subjects who have an Hgb level of more than 13.0 g/dL and number of episodes will be summarized. On-therapy Hgb values observed in both scheduled and unscheduled visits will be included in the summary. This will be also summarized by baseline dialysis status.

#### Scatter plot of Hgb assessments: Central Laboratory vs. HemoCue

A scatter plot of Hgb values measured by Central Laboratory versus Hgb values measured by Hemocue will be produced along with Pearson's correlation coefficient. All available pairs of Hgb (i.e. non-missing values in both from central laboratory and from the corresponding HemoCue measurement) will be used.

#### Iron Use

#### Dose of i.v. iron during the treatment period

Average quarterly i.v. iron dose (See Section 10.6.3) will be summarized using mean, standard deviation, minimum, P25, median, P75, and maximum. Quarter 1 (Day 1 to Week 12) and Quarter 2 (Week 12 to Week 24) will be used. This will be also summarized by baseline dialysis status.

#### Number (%) of subjects who use iron during the treatment period

The number and percentage of subjects who use iron (both i.v. and oral iron) during the treatment period will be summarized. This will be also summarized by baseline dialysis status.

#### • Iron Parameter (ferritin, TSAT, hepcidin, serum iron, and TIBC)

Based on literature review the distributions of TSAT and hepcidin are skewed and require a log-transformation (See Section 10.6.3).

#### Raw observed value at each assessment visit

Ferritin, serum iron, and TIBC values will be summarized using mean, standard deviation, 95%CI, minimum, P25, median, P75, and maximum at each assessment visit. TSAT and hepcidin values will be summarized using geometric mean, standard error, coefficient of

variation, and 95%CI based on log-transformed parameters, and median, minimum, and maximum based on original scale at each assessment visit. This will be also summarized by baseline dialysis status.

#### Change from baseline at each assessment visit

Change from baseline in Ferritin, serum iron, and TIBC values will be summarized using mean, standard deviation, 95%CI, minimum, P25, median, P75, and maximum at each assessment visit. Percent Change from baseline in TSAT and hepcidin values will be summarized using geometric mean and 95%CI based on log-transformed parameters, and median, minimum, and maximum based on original scale at each assessment visit. Graphical summaries will be provided using mean and 95% CI over time. This will be also summarized by baseline dialysis status.

#### • Dose adjustment

The dose adjustment algorithm is described in Section 10.6.3, based on HemoCue Hgb values including those in both scheduled and unscheduled visits

#### Dose level (mg) at each assessment visit

The values will be summarized using mean, standard deviation, minimum, P25, median, P75, mode, and maximum at each assessment visit. The mean dose during Week 12 to 24 will also be summarized. This will be also summarized by baseline dialysis status.

#### Duration (days) of treatment interruption due to Hgb >13.0 g/dL

The number and percentage of subjects who have a period of treatment interruption due to Hgb >13.0 g/dL will be summarized. On subjects who have a period of treatment interruption due to Hgb >13.0 g/dL, the duration (in days) of treatment interruption due to Hgb >13.0 g/dL per subject will be summarized using mean, standard deviation, minimum, P25, median, P75, and maximum. Hgb values observed in both scheduled and unscheduled visits will be counted in the summary. This will be also summarized by baseline dialysis status.

#### Dose adjustment

The number and percentage of subjects with dose adjustments will be provided. Number of dose adjustments will be summarized using mean, standard deviation, minimum, median, mode, and maximum. For dose adjustments frequency, the number and percentage of subjects will be provided by the number of dose adjustments (i.e. zero, one, two, three, four, and five or more). For timing of dose adjustments, the number and percentage of subjects with dose adjustments by each assessment visit will be provided. This will be also summarized by baseline dialysis status.

Number (%) of subjects with each dose level at each assessment visit

The number and percentage of subjects with each dose level adjustments will be provided. Graphical summaries will be provided with the number of subjects in each dose level. Dose level categories will be classified into 10; W/d (early withdrawal), 0 mg (treatment interruption), 1 mg, 2 mg, 4 mg, 6 mg, 8 mg, 12 mg, 18 mg, and 24 mg). This will be also summarized by baseline dialysis status.

#### Number of dose adjustment to reach the lower Hgb target (10.0 g/dL)

The number and percentage of subjects with dose adjustments to reach the lower Hgb target will be provided on the basis of on-therapy Hgb. Number of dose adjustment to reach the lower Hgb target will be summarized using mean, standard deviation, minimum, median, mode, and maximum. For dose adjustments frequency, the number and percentage of subjects will be provided by the number of dose adjustments (i.e., zero, one, two, three, four, five or more). Subjects who does not reach the lower Hgb target during treatment period will be excluded from the summary. This will be also summarized by baseline dialysis status.

#### Other

The following two sorts of scatter plots of interest will be produced for overall and dialysis status groups:

Change from baseline in Hgb at Week 4 versus the candidate covariates

Mean dose during Week 12 to 24 versus the candidate covariates

See Appendix 10 for the candidate covariates and Section 10.6.3 for the detailed derivations.

#### 8.1.3. Planned Hgb Efficacy Statistical Analyses

#### **Secondary Hgb Analyses**

#### Endpoint(s)

- Hgb and changes from baseline
- Number (%) of subjects who have a Hgb level within the target range (10.0–12.0 g/dL)
- Time (in days) to reach the lower target Hgb level (10.0 g/dL)
- Number (%) of subjects who have a Hgb level of less than 7.5 g/dL
- Number (%) of subjects who have a Hgb increase of more than 2.0 g/dL over any 4 weeks
- Number (%) of subjects who have a Hgb level of more than 13.0 g/dL and number of episodes

#### **Model Specification**

- Hgb values from central laboratory will be used, unless otherwise specified. However, if a
  central laboratory Hgb value is missing, a corresponding non-missing HemoCue Hgb value will
  be used (See Section 10.6.3).
- The secondary analysis is to assess appropriate control of Hgb within the target range, on the basis of the Hgb mean at Week 24 and the number (%) of subjects with Hgb within the target

#### **Secondary Hgb Analyses**

range as secondary endpoints.

- For the Hgb, the summary statistics will be calculated, along with the two-sided 95% confidence interval based on t-distribution.
- The percentage of subjects with Hgb within the target range will be calculated at Week 24, with calculation of exact two-sided 95% confidence interval based on binomial distribution.
- The time (in days) to reach first the lower target Hgb level (10.0 g/dL) will be calculated in each subject, and summarized descriptively by Kaplan-Meier method using P25, median, and P75.
   Subjects who could not reach lower target will be regarded as censored at Study Treatment Stop Date (See Section 10.6.1).

#### 8.2. Safety Analyses

The safety analyses will be based on the All Treated Subjects population, unless otherwise specified.

Table 5, Table 6, and Table 7 provide overviews of the planned analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

#### 8.2.1. Overview of Planned Adverse Events Analyses

All AEs will be categorized by the MedDRA (version 20.0 or higher if available) system organ class and preferred term to tabulate the number and incidence.

AEs of special interest will be manually-selected at patient-level (i.e. following case-by-case review by members of the SRT including representatives from the local Japan team) and not at preferred term level.

Table 5 Overview of Planned AEs Analyses

| Endpoint / Parameter/ Display Type | | Absol | olute |
|---|---|---|---|
| | Sun | nmary | Individual |
| | T | F | L |
| Adverse Events (AEs) | | | |
| On-therapy AEs by SOC and PT | Υ | | Υ |
| On-therapy AEs by SOC and PT | Υ | | |
| by Dialysis Status | I | | |
| On-therapy AEs by SOC and PT and Maximum Intensity | Υ | | |
| On-therapy AEs up to Week 4 by SOC and PT | Υ | | |
| On-therapy AEs up to Week 4 by SOC and PT | Υ | | |
| by Dialysis Status | ī | | |
| On-therapy AEs up to Week 4 by SOC and PT and Maximum Intensity | Υ | | |
| Post-therapy AEs by SOC and PT | Y | | Υ |
| Post-therapy AEs by SOC and PT and Maximum Intensity | Y | | |
| On-therapy Drug-Related AEs by SOC and PT | Υ | | |
| On-therapy Drug-Related AEs by SOC and PT | Υ | | |
| by Dialysis Status | ľ | | |
| On-therapy Drug-Related AEs by SOC and PT and Maximum Intensity | Y | | |
| On-therapy Drug-Related AEs up to Week 4 by SOC and PT | Y | | |
| On-therapy Drug-Related AEs up to Week 4 by SOC and PT | Υ | | |
| by Dialysis Status | Y | | |
| On-therapy Drug-Related AEs up to Week 4 by SOC and PT and Maximum | Υ | | |
| Intensity | Ť | | |
| Post-therapy Drug-Related AEs by SOC and PT | Υ | | |
| Post-therapy Drug-Related AEs by SOC and PT and Maximum Intensity | Y | | |
| On-therapy Common (>= 5 %) Non-Serious AEs by SOC and PT (Subjects & | Υ | | |
| No. of Occurrences) | ' | | |

| Endpoint / Parameter/ Display Type | | Absol | lute |
|---|---|---|---|
| | Sun | nmary | Individual |
| | Т | F | L |
| Subject Numbers for Individual AEs | | | Υ |
| Relationship Between AE SOCs, PT & Verbatim Text | | | Υ |
| Serious and Other Significant AEs | | | |
| Fatal Serious AEs | | | Υ |
| Non-Fatal Serious AEs | | | Υ |
| On-therapy Serious AEs | Υ | | |
| Post-therapy Serious AEs | Υ | | |
| Serious AEs in Screening Period [1] | | | Υ |
| Reasons for Considering as a Serious AE | | | Υ |
| Serious AEs by SOC and PT (Subjects & No. of Occurrences) | Υ | | |
| AEs Leading to Withdrawal from Study / Permanent Discontinuation of Study | Υ | | Υ |
| Treatment by SOC and PT | ' | | ' |
| CV Events | | | Υ |
| AEs of special interest [2] | | | |
| On-therapy AEs of special interest | Υ | | Υ |
| On-therapy AEs of special interest | Υ | | |
| by Dialysis Status | · · | | |
| Post-therapy AEs of special interest | Υ | | Υ |
| Other Safety Summary for Plain Language Summary | | | |
| On-therapy Serious Drug-Related AEs | Υ | | |
| On-therapy Non-Serious Drug-Related AEs | Υ | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Listing will be based on All Screening Population.
- [2] See Section 10.6.4.

#### 8.2.1.1. Planed AE Analyses Displays

#### Adverse Events

#### AEs by SOC and PT

The number and percentage of subjects reporting at least one AE will be provided. These events will be summarized by primary system organ class and preferred term. On-therapy, on-therapy up to week 4, and post-therapy AEs will be summarized separately. On-therapy AE will be also summarized by baseline dialysis status.

#### AEs by SOC and PT and Maximum Intensity

AEs will be summarized by Maximum Intensity (not applicable, mild, moderate, or severe) by primary system organ class and preferred term. Subjects who experience the same event several times with different intensities will only be counted with the maximum intensity in the order of (not applicable < mild < moderate < severe). Ontherapy, on-therapy up to week 4, and post-therapy AEs will be summarized separately.

#### Drug-Related AEs by SOC and PT

The number and percentage of subjects reporting at least one drug-related AE will be provided. These events will be summarized by primary system organ class and preferred term. On-therapy, on-therapy up to week 4, and post-therapy AEs will be summarized separately. On-therapy AE will be also summarized by baseline dialysis status.

#### Drug-Related AEs by SOC and PT and Maximum Intensity

Drug-related AEs will be summarized by Maximum Intensity (not applicable, mild, moderate, or severe) by primary system organ class and preferred term. Subjects who experience the same event several times with different intensities will only be counted with the maximum intensity in the order of (not applicable < mild < moderate < severe). On-therapy, on-therapy up to week 4, and post-therapy AEs will be summarized separately.

## On-therapy Common (>= 5 %) Non-Serious AEs by SOC and PT (Subjects & No. of Occurrences)

The number and percentage of subjects reporting at least one on-therapy common ( $\geq$  5 %) non-serious AE will be provided. The number of on-therapy non-serious AE occurrences will also be provided. These events will be summarized by primary system organ class and preferred term.

#### • Serious and Other Significant AEs

#### Serious AEs

The number and percentage of subjects reporting at least one Serious AE will be provided. These events will be summarized by primary system organ class and preferred term. On-and post-therapy serious AEs will be summarized separately.

#### On-therapy Serious AEs by SOC and PT (Subjects & No. of Occurrences)

The number and percentage of subjects reporting at least one on-therapy serious AE will be provided. The number of on-therapy serious AE occurrences will also be provided. These events will be summarized by preferred term.

<u>AEs Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment</u> by SOC and PT The number and percentage of subjects reporting each on-therapy AE leading to discontinuation of study treatment will be summarized. These events will be summarized by preferred term.

#### • AEs of Special Interest (AESIs)

How to identify the AESIs is described in Section 10.6.4.

#### AEs of Special Interest

The number and percentage of subjects reporting at least one AESI will be provided. These events will be summarized by each AESI term (See Section 10.6.4). On-therapy and post-therapy AESIs will be summarized separately. On-therapy AE will be also summarized by baseline dialysis status.

#### • Other Safety Summary for Plain Language Summary

#### Serious/Non-serious Drug-Related AEs

The number and percentage of subjects with on-therapy serious or non-serious drugrelated AEs will be summarized by preferred term. The serious AEs and the non-serious AEs will be summarized separately.

#### 8.2.2. Overview of Planned Clinical Laboratory Analyses

Table 6 Overview of Planned Clinical Laboratory Analyses

| Endpoint / Parameter/ Display Type | | Abs | bsolute Change | | | from BL |
|---|---|---|---|---|---|---|
| | Sum | mary | Individual | Sumr | nary | Individual |
| | Т | F | L | Т | F | L |
| Chemistry | | | | | | |
| Chemistry Values by Visit | Υ | | Υ | Υ | | |
| Percent change from Baseline in Lipid Parameters [1] (total cholesterol, LDL cholesterol, and HDL cholesterol) | | | Y | Υ | Υ | |
| Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline | Υ | | | | | |
| Worst Case Chemistry Results Relative to PCI Criteria Post-Baseline Relative to Baseline | Υ | | | | | |
| Hematology | | | | | | |
| Hematology Values by Visit | Υ | | Υ | Υ | | |
| Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline | Υ | | | | | |
| Worst Case Hematology Results Relative to PCI Criteria Post-Baseline Relative to Baseline | Υ | | | | | |
| Other Laboratory Tests [2] | | | | | • | |

| Endpoint / Parameter/ Display Type | Absolute | | | Ch | ange | from BL |
|---|---|---|---|---|---|---|
| | Summary | | Individual | Summary | | Individual |
| | T | F | L | Т | F | L |
| Other Laboratory Values by Visit [2] | Υ | | Υ | Υ | | |
| Worst Case Other Laboratory Results Relative to Normal Range Post-Baseline Relative to Baseline [2] | Υ | | | | | |
| Worst Case Other Laboratory Results Relative to PCI Criteria Post-Baseline Relative to Baseline [2] | Υ | | | | | |
| Hepatobiliary (Liver) | | | | | | |
| Liver Monitoring/Stopping Event Reporting | Υ | | | | | |
| Hepatobiliary Laboratory Abnormalities | Υ | | | | | |
| Medical Conditions for Subjects with Liver Stopping Events | | | Y | | | |
| Substance Use for Subjects with Liver Stopping Events | | | Υ | | | |
| Scatter Plot of Maximum vs. Baseline for ALT | | <b>Y</b> [3] | | | | |
| Scatter Plot of Maximum ALT vs Maximum Total Bilirubin | | <b>Y</b> [3] | | | | |
| All Laboratory | | | | | | |
| All Laboratory Data for Subjects with any Value of Potential Clinical Concern/PCI | | | Y | | | |
| Laboratory Values of PCI | | | Υ | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Lipid parameters will be log-transformed and the percent change from baseline will be reported.
- [2] Only iPTH will be collected as other laboratory tests.
- [3] This figure may not be provided in this study because this is required for 'larger study' by the GSK Core RAP requirements in the RAP Template.

#### 8.2.2.1. Planned Clinical Laboratory Analyses Displays

#### • Chemistry/Hematology/Other Laboratory Tests

#### Clinical Laboratory Values by Visit

The values will be summarized using mean, standard deviation, median, minimum, and maximum at each assessment visit and baseline. Chemistry values, hematology values, and other laboratory values will be summarized separately.

#### <u>Percent change from Baseline in Lipid Parameters</u>

Lipid parameters will be log-transformed and the percent change from baseline will be reported. The percent change from baseline in each lipid parameter, including baseline values, will be summarized using geometric mean, 95% CI, minimum, median, and maximum at each assessment visit. In baseline values, the coefficient of variation will also be provided.

#### Clinical Laboratory Changes from Baseline by Visit

The values will be summarized using mean, standard deviation, median, minimum, and maximum at each assessment visit. Change from baseline in chemistry, hematology, and other laboratory will be summarized separately.

<u>Worst Case Laboratory Results Relative to Normal Range/PCI Criteria Post-Baseline</u> Relative to Baseline

The number of subjects with worst laboratory results relative to normal range/potential clinical importance (PCI) criteria which are post-baseline relative to baseline, including unscheduled assessments, will be summarized by test and category. Summaries for normal range and PCI will be provided separately. The categories for normal range are: To Low, To Normal or No Change, To High; the categories for PCI criteria are: To Low, To w/in Range or No Change, To High. The categorization is determined by comparing the baseline category to the worst case post-baseline category.

#### • Hepatobiliary (Liver)

Details of liver chemistry stopping criteria are described in the protocol.

Liver monitoring/stopping events will be summarized.

Hepatobiliary laboratory abnormalities will be summarized.

A scatter plot of maximum on-therapy ALT values versus baseline ALT values will be produced if larger data permit.

A scatter plot of maximum total bilirubin (xULN) versus maximum ALT (xULN) values on-therapy will be produced if larger data permit.

#### 8.2.3. Overview of Planned Other Safety Analyses

Table 7 Overview of Planned Other Safety Analyses

| Endpoint / Parameter/ Display Type | | Absolute | | | ange | from BL |
|---|---|---|---|---|---|---|
| | Sum | mary | Individual | Sumr | nary | Individual |
| | Т | F | L | Т | F | L |
| ECG | | | | | | |
| ECG Findings by Visit | Υ | | Υ | | | |
| ECG Values by Visit | | | Υ | Υ | | |
| Abnormal ECG Findings | | | Υ | | | |
| Vital Signs | | | | | | |
| Vital Signs by Visit | Υ | | Υ | Υ | | |
| Worst Case Vital Sign Results Relative to PCI Criteria Post-Baseline Relative to Baseline | Υ | | | | | |

| Endpoint / Parameter/ Display Type | Absolute | | | Cha | from BL | |
|---|---|---|---|---|---|---|
| | Summary | | Individual | Sumn | nary | Individual |
| | Т | F | L | Т | F | L |
| All Vital Signs for Subjects with Values of PCI | | | Υ | | | |
| Ophthalmology | | | | | | |
| Ophthalmologic Exams at Screening | Υ | | Y | | | |
| On-Therapy Ophthalmologic Exams | Υ | | Υ | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8.2.3.1. Planned Other Safety Analyses Displays

#### ECG

ECG findings ('normal', 'abnormal, not clinically significant', 'abnormal, clinically significant') will be summarized by each assessment visit. Findings without regard to visits (labelled "Worst Case Post-Baseline", only the worst case finding for each subject, will also be provided. All ECG measures (heart rate, PR interval, QRS duration, QT (uncorrected) interval and QTcB (calculated), result of ECG) will be included in a subject listing.

#### • Vital Signs

Vital sign values will be summarized using mean, standard deviation, minimum, median, and maximum for each assessment visit. Separate summary statistics of pre- and post-dialysis vital signs will be provided for raw values and change from baseline. In a summary of change from baseline, each baseline value (i.e. pre- and post-dialysis baseline) will be used for calculation (Section 10.5.2).

The number of subjects with worst case vital sign results relative to PCI criteria which are post-baseline relative to baseline, including unscheduled assessments, will also be summarized by test and category. The categories for PCI criteria are: To Low, To w/in Range or No Change, To High. The categorization is determined by comparing the baseline category to the worst case post-baseline category.

#### • Ophthalmology Exams

The responses to each question will be summarized using number and percentage at each assessment visit. The response will be classified into 'Yes' and 'No'. Ophthalmology exam at screening and at on-therapy will be summarized separately. The number of subjects with worst case after-screening ophthalmology exams (i.e., the response is 'Yes' at least once during whole treatment period, including unscheduled visits) will also be summarized by each question.

#### 8.3. Pharmacokinetic Analyses

#### 8.3.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the PK population, unless otherwise specified.

Table 8 provides an overview of the planned analyses, with full details being presented in Appendix 14: List of Data Displays. Summaries will be produced for week 12, week 24, and pooled.

Table 8 Overview of Planned Pharmacokinetic Analyses

| Endpoints | Untransformed | | | | Log-Transformed | | | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Individual | | Summary | | Individual | |
| | F | T | F | L | F | T | F | L |
| Plasma Concentrations of GSK1278863 | Y [1] [2] | Y | Υ [1] | Y | | | | |
| Derived PK Parameters | <b>Y</b> [3] | <b>Y</b> [3] | <b>Y</b> [3] | Υ | | Υ[3] | | |
| Dose Normalized PK<br>Parameters | <b>Y</b> [3] | <b>Y</b> [3] | <b>Y</b> [3] | Y | | <b>Y</b> [3] | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Linear and Semi-Log plots will be created on the same display.
- 2. Separate Mean (± SD) and Median plots will be generated.
- 3. Individual PK parameters calculated less than 4 time point concentration or any time deviated concentration will be omitted from summaries and figures.

#### 8.3.2. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Process & Standards).

Concentrations of GSK1278863 in plasma will be listed and summarized by dose group and nominal time. Individual plasma concentration-time profiles and median/mean profiles by dose group will be plotted. Each of figures will contain one plot on the untransformed scale (i.e. a linear plot) and one plot on the log transformed scale (i.e. a log-linear plot).
#### 8.3.3. Pharmacokinetic Parameters

#### 8.3.3.1. Deriving Pharmacokinetic Parameters

- Derivation of pharmacokinetic parameters will be performed by, or under the direct auspices of, Clinical Pharmacology & Science Promotion Office, GlaxoSmithKline K.K.
- Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using Win Nonlin (version 6.3 or higher).
- All calculations of non-compartmental parameters will be based on actual sampling times.
- Pharmacokinetic parameters described in Table 9 will be determined from the Plasma GSK1278863 concentration-time data, as data permits.

Table 9 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-4) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(last)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the linear trapezoidal for each decremental trapezoid. The concentration at 0 hr will be set to 0. |
| AUC(0-7) | Area under the concentration-time curve from time zero to seven will be calculated using the linear trapezoidal rule for each incremental trapezoid and the linear trapezoidal for each decremental trapezoid. The concentration at 0 hr and 7 hr will be set to 0. |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| Tmax | Time to first occurrence of Cmax will be obtained directly from the concentration-time data. |

#### NOTES:

- Additional parameters may be included as required.
- C(last) is expected to be the concentration observed at 4hours after the most recent dose.

#### 8.3.4. Population Pharmacokinetic (PopPK) Analyses

No population pharmacokinetic analysis is planned.

## 8.4. Pharmacodynamic Analyses

No pharmacodynamic analysis is planned.

## 8.5. Pharmacokinetic / Pharmacodynamic Analyses

No pharmacokinetic / pharmacodynamic analysis is planned.


204716

## 9. REFERENCES

N/A

## 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| RAP Section 5 | General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.2 | Appendix 2: Time and Events |
| Section 10.3 | Appendix 3: Assessment Windows |
| Section 10.4 | Appendix 4: Treatment States & Phases |
| Section 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| | <ul> <li>Study Treatment &amp; Sub-group Display Descriptors</li> </ul> |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.6 | Appendix 6: Derived and Transformed Data |
| | General, Study Population & Safety |
| | • Efficacy |
| | Pharmacokinetic |
| Section 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 10.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 10.9 | Appendix 9: Multicenter Studies |
| | Laboratory Values |
| | • ECG |
| | Vital Signs |
| Section 10.10 | Appendix 10: Examination of Covariates and Subgroups |
| Section 10.11 | Appendix 11: Multiple Comparisons and Multiplicity |
| Section 10.12 | Appendix 12: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | endices |
| Section 10.13 | Appendix 13: Abbreviations & Trade Marks |
| Section 10.14 | Appendix 14: List of Data Displays |
| Section 10.15 | Appendix 15: Example Mock Shells for Data Displays |

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

Per Protocol Population will not be defined in this study.

## 10.2. Appendix 2: Time & Events

## 10.2.1. Protocol Defined Time & Events

| Period | Scre | ening | | | | Trea | tment | | | | Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visits All assessments pre-dialysis, unless noted. | | Week<br>-4 | Day 1 | Week<br>4 | Week<br>8 | Week<br>12 | Week<br>16 | Week<br>20 | Week<br>24 | Early<br>withdraw<br>al <sup>10</sup> | 2–4 weeks<br>after Week 24<br>or early<br>withdrawal |
| Allowable window (days) | | ±7 | - | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | - | ±3 |
| Informed consent | X | | | | | | | | | | |
| Inclusion/exclusion | | X | X | | | | | | | | |
| Medical history, demography, height, body weight <sup>1</sup> | | X | | | | | | | | | |
| IWRS call | | X | X | X | X | X | X | X | X | X | X |
| Study medication dispensing <sup>2</sup> | | | X | X | X | X | X | X | | | |
| Study medication compliance | | | | X | X | X | X | X | X | X | |
| Vital signs (before and after dialysis) <sup>3</sup> | | X | X | X | | X | | | X | X | X |
| Ophthalmology examination <sup>4</sup> | | X 11 | | | • | <b>→</b> | | <b>←</b> | | <b>←→</b> | |
| ECG | | X | | | | X | | | X | | |
| HemoCue Hgb | | | X | X | X | X | X | X | X | | |
| Hematology | | X 12 | X | X | Hgb<br>only | X | Hgb<br>only | Hgb<br>only | X | X | X |
| Clinical chemistry | | X | X | X | | X | | | X | X | X |
| Ferritin, TSAT | | X | X | X | | X | | | X | X | |
| Serum iron, TIBC, UIBC, serum transferrin, hepcidin | | | X | X | | X | | | X | X | |
| Serum pregnancy test <sup>5</sup> | | X | X | X | | X | | | X | X | X |
| Estradiol <sup>5</sup> , FSH <sup>6</sup> | | X | | | | | | | | | |
| Pharmacokinetics <sup>7</sup> | | | | | | X | | | X | | |
| iPTH | | | X | X | | X | | | X | | |
| Genetics sample <sup>8</sup> | | | X | | | | | | | | |
| Adverse event assessment 9 | | | - | | | | <b>→</b> | | | | |
| Concomitant medication assessment | | <b>—</b> | <u> </u> | <u> </u> | | <b>—</b> | | | | | |

- 1. Body weight is measured after dialysis.
- 2. If a subject visit the study site only to receive study medication, only the IWRS call, study medication dispensing, and study medication compliance will be required
- 3. At visits without dialysis, only one measurement of each parameter will be obtained.
- 4. Ophthalmology exams should be conducted at the following time points.
  - Screening: anytime after consenting and prior to first dose of study medication (Day 1)
  - Week 12: window from weeks 10-14 (inclusive)
  - End of study: window from weeks 20-24 (inclusive)
  - Early study medication discontinuation or study withdrawal: withdrawal eye exam as close to the last dose as possible.
     Re-conduct is not required if the exam is conducted within two weeks prior to withdrawal visit.
- 5. Only for females of reproductive potential.
- 6. Only at determination of menopausal status in female subjects (Section 5.1).
- 7. See Table 7
- 8. For optional genetic research, informed consent should be obtained before the specimen collection.
- See Section 7.4.1.
- 10. For examination at early withdrawal, the specified assessments should be performed as far as possible
- 11. The previous result of ophthalmology exam at the screening may be used if the subject meets all of the following criteria and the investigator judges it appropriate.
  - There were no findings that would suggest a repeat ophthalmology exam performed within the next 3 months at the latest screening ophthalmology exam.
  - Subjects had no new eye-related symptoms or complaints since the latest screening ophthalmology exam.
  - The latest screening ophthalmology exam was performed within 3 months prior to anticipated Day 1.
- 12. Exam should be conducted at least one week after ESA treatment

#### • Blood Sampling Schedule for Pharmacokinetics

| PK sample | Week 12 <sup>2</sup> | Week 24 <sup>2</sup> |
|---|---|---|
| Blood sampling timing <sup>1</sup> | 1, 2, 3, and 4 h after a | administration of GSK1278863 |

Subjects must take the study medication in consideration of blood sampling time. Subjects will record the date and time of the last two study medication doses taken prior to blood sampling in the medication diary. Preferably, there should be an interval of at least 12 h between these two doses.

- 1. Blood sampling should be completed within +/- 30 min of the planned collected time.
- 2. Blood sampling not performed at this visit may be postponed until the following visits.

#### 10.3. Appendix 3: Assessment Windows

All data will be reported according to the nominal visit date for which it was reported (that is, no visit windows will be applied during dataset creation). Permissible range at each visit was specified in time & event table (See Appendix 2). Records in the eCRF unscheduled visit will not be slotted to a particular time point, but remain as unscheduled if they are either summarized or listed unless otherwise specified.

#### 10.3.1. Definitions of Analysis Time Point

| Analysis Time Point | Definitions |
|---------------------|-----------------------------------|
| Screening [1] | Data collected in Screening visit |
| Day 1 [1] | Data collected in Day 1 visit |
| Week 4 | Data collected in Week 4 visit |
| Week 8 | Data collected in Week 8 visit |
| Week 12 | Data collected in Week 12 visit |
| Week 16 | Data collected in Week 16 visit |
| Week 20 | Data collected in Week 20 visit |
| Week 24 | Data collected in Week 24 visit |
| Follow-up | Data collected in Follow-up visit |

Note: Any unscheduled visit will not be slotted to a particular time point.

<sup>[1]</sup> For rescreened subjects, data collected in screening-pass visit will be used for analysis. They may have multiple records at Screening and/or Day 1 visit, which associates with a screening-pass visit and screening failure visit(s)

### 10.4. Appendix 4: Treatment States and Phases

#### 10.4.1. Treatment States

Assessments and events will be classified according to time of occurrence relative to the randomization date and study treatment stop date.

#### 10.4.1.1. Treatment States for Hgb Data

| Treatment State | Definition |
|---|---|
| Pre-therapy | Date ≤ Randomization Date |
| On-therapy | Randomization Date < Date ≤ Study Treatment Stop Date + 1 day |
| Post-therapy | Date > Study Treatment Stop Date + 1 day |

#### NOTES:

- If Randomization date is missing then the assessment will be consider to be Pre-therapy
- If study treatment stop date is missing then the assessment will be considered to be On-therapy

#### 10.4.1.2. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-therapy | AE Start Date < Randomization Date |
| On-therapy | If AE onset date is on or after randomization date & on or before Study Treatment Stop Date + 1 day |
| | Randomization Date ≤ AE Start Date ≤ Study Treatment Stop Date + 1 day |
| Post-therapy | If AE onset date is after Study Treatment Stop Date + 1 day |
| | AE Start Date > Study Treatment Stop Date + 1 day |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 day |
| Drug-related | If relationship is marked 'YES' on eCRF or value is missing. |

#### NOTES:

- If Randomization date is missing then the assessment will be consider to be Pre-therapy
- If study treatment stop date is missing then the AE will be considered to be On-therapy.

#### 10.4.1.3. Treatment States for Concomitant Medications Data

| Treatment State | Definition |
|---|---|
| Pre-therapy | Concomitant Medication Start Date ≤ Randomization Date |
| On-therapy | Define as (A) or (B) |
| | (A): If concomitant medication start date is on or after randomization date & on or before Study Treatment Stop Date |
| | • Randomization Date ≤ Concomitant Medication Start Date ≤ Study Treatment Stop Date |
| | If Study Treatment Stop Date is missing, just check if the start date is on or after randomization date. (B): If concomitant medication start date is before randomization date & concomitant medication stop date is on or after randomization date |
| | Concomitant Medication Start Date < Randomization Date |

| Treatment State | Definition |
|---|---|
| | Randomization Date ≤ Concomitant Medication Stop Date |
| Post-therapy | Concomitant Medication Stop Date > Study Treatment Stop Date |
| | If Study Treatment Stop Date is missing: |
| | post-therapy = blank |
| | where Concomitant Medication Stop Date ≥ Randomization Date |
| | post-therapy = Y |
| | where concomitant medication stop date are missing |
| | <ul><li>post-therapy = N</li></ul> |
| | where Concomitant Medication Stop Date < Randomization Date |

#### NOTES:

- If Randomization date is missing then the assessment will be consider to be Pre-therapy
- Data of concomitant medication includes ESA, iron, and blood products and blood supportive care products.

Illustrations of the pre-therapy, on-therapy, and post-therapy treatment states for concomitant medications are included below:

| | Pre-<br>therapy | On-therapy | | Pos | st-therapy | Pre-therapy medication | On-therapy medication | Post-therapy medication | |
|---|---|---|---|---|---|---|---|---|---|
| (a) | хх | | | | /s | | Υ | N | N |
| (b) | x | | ——х | - | Days | | Υ | Υ | N |
| (c) | x | | | Study Treatment Stop Date | +1 | ——х | Υ | Υ | Υ |
| (d) | | Randomization Date | xx | ] dc | ate . | | N | Υ | N |
| (e) | | u [ | х | Stc | Study Treatment Stop Date | ———х | N | Υ | Y |
| (f) | | atic | | ent | top | хх | N | N | Y |
| (g) | ?x | niz | | Ţ. | ıt S | | Υ | N | N |
| (h) | ? | do | ——х | -g | mel | | Y* | Υ | N |
| (i) | ? | Ran | | <u> </u> | eat | ———х | Y* | Y* | Υ |
| (j) | X | - | | ğ | Ĕ | ? | Υ | Y** | Y** |
| (k) | | | х | 0, | ud | <del>?</del> | N | Υ | Y** |
| (l) | | | | | Sţ | x? | N | N | Y |
| (m) | ?——— | | | | | <del>?</del> | Y*** | Y*** | Y*** |
| (n) | х | Х | | | | | Υ | Υ | N |
| (o) | ?——— | Х | | | | | Y* | Υ | N |
| (p) | | Х | ——х | | | | N | Υ | N |
| (q) | | Х | | Χ | | | N | Υ | N |
| (r) | | | | Χ | _ | ———Х | N | Υ | Y |
| (s) | | | | Χ | _ | <del>?</del> | N | Υ | Y** |
| (t) | | | | | Χ | ———Х | N | N | Y |
| (u) | | | | | Χ | <del>?</del> | N | N | Y |
| (v) | | | x | _ | Χ | | N | Υ | Y |

x = start/stop date of medication

<sup>? =</sup> missing start/stop date of medication

<sup>\*</sup> If a medication is stopped On-therapy or Post-therapy and no start date is recorded it will be assumed that the medication was ongoing from the Pre-therapy phase

<sup>\*\*</sup> If a medication is started Pre-therapy or On-therapy and no stop date is recorded then usage will be assumed to be ongoing for the remainder of the study

<sup>\*\*\*</sup> If a medication has no start or stop date it will be assumed that the medication was ongoing from the Pretherapy phase to the Post-therapy phase

## 10.5. Appendix 5: Data Display Standards & Handling Conventions

#### 10.5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Reporting | |
| Code | Description | Description | Order |
| D1 | GSK1278863 | GSK1278863 | 1 |

#### 10.5.2. Baseline Definition & Derivations

#### 10.5.2.1. Baseline Definitions

The baseline value will be the latest pre-dose assessment. This is generally expected to be the pre-dose value from the Day 1 visit, except for ECG. For ECG, screening assessment will be used as a baseline.

For vital signs, the baseline value at pre- and post-dialysis will be defined differently.

#### 10.5.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| Change from Baseline<br>For Vital Signs | <ul> <li>Pre-dialysis: <ul> <li>Post-Dose Visit Value from Pre-Dialysis Assessment –</li> <li>Baseline from Pre-Dialysis Assessment</li> </ul> </li> <li>Post-dialysis: <ul> <li>Post-Dose Visit Value from Post-Dialysis Assessment –</li> <li>Baseline from Post-Dialysis Assessment</li> </ul> </li> </ul> |
| % Change from Baseline<br>For TSAT, Hepcidin, and Lipid<br>Parameters | <ol> <li>Log-transform the data at both the baseline and the specified timepoint</li> <li>Calculate a change from baseline using the log-transformed data for each subject</li> <li>Calculate the mean, and 95%CI and standard error (SE) of the log-transformed data</li> <li>Exponentially back-transform to the original scale</li> <li>Subtract 1, then multiply everything by 100%</li> <li>So, geometric mean for percent change from baseline = { exp(Mean [ln(Post-Dose Visit Value) - ln(Baseline)]) - 1 }x</li> </ol> |

| Definition | Reporting Details |
|------------|----------------------------------------------------------------|
| | Coefficient of variation will be calculated as |
| | CV%=[exp(Var in log scale)-1 ] <sup>1/2</sup> x 100 |
| | where 'Var in log scale' represents variance of percent change |
| | from baseline in log scale. |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.5.2.1 will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing, no derivation will be performed and will be set to missing.

#### 10.5.3. Reporting Process & Standards

| Reporting Process | Reporting Process |
|---|---|
| Software | |
| The currently su | The currently supported versions of SAS software and S-Plus will be used. |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Area | : /arenv/arprod/gsk1278863/mid204716/final_01 |
| QC Spreadsheet | : /arenv/arprod/gsk1278863/mid204716/final_01/documents |
| <b>Analysis Datasets</b> | Analysis Datasets |
| Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.1.3 & ADaM IG Version 1.0. For creation of ADaM datasets (ADCM/ADAE), the same version of distingery datasets will be | |
| • For creation of | ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be |

#### Generation of RTF Files

Not generated.

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - o 4.03 to 4.23: General Principles
  - o 5.01 to 5.08: Principles Related to Data Listings
  - o 6.01 to 6.11: Principles Related to Summary Tables
  - o 7.01 to 7.13: Principles Related to Graphics

implemented for conversion from SI to SDTM.

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.

#### **Planned and Actual Time**

#### **Reporting Standards**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - For Individual PK figures, the plot will use actual relative time.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Scheduled visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings, figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables, unless otherwise specified.
  - If unscheduled visits are included in a summary, it will be provided how a summary will be produced as appropriate.
- Unscheduled visits will not be included in figures, unless otherwise specified.
- All unscheduled visits will be included in listings.

Refer to IDSL Statistical Principals 7.01 to 7.13.

| Descriptive Summa | ry Statistics |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1: This does not apply to the output of statistical models or when the standard list is inappropriate. |
| | <ul> <li>Hgb and iron summary statistics will include 95%Cl and percentiles (F<br/>and P75).</li> </ul> |
| | Dose level and dose adjustment frequency summary statistics will include mode. |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharm | acokinetic Concentration Data |
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Reporting of Pharm | acokinetic Parameters |
| Descriptive<br>Summary Statistics<br>(Log Transformed) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of log-transformed data and between geometric coefficient of variation (CVb (%)) will be reported. [1] CV <sub>b</sub> (%) = √ (exp(SD²) - 1) * 100 (SD = SD of log transformed data) |
| <b>Graphical Displays</b> | ( |

### 10.6. Appendix 6: Derived and Transformed Data

#### 10.6.1. General

#### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.
- For multiple measurements at Screening and Day 1 visit, the screening-pass visit record will be used for analysis (See Appendix 3).

#### **Study Day**

- Calculated as the number of days from randomization date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Randomization Date → Study Day = Ref Date Randomization Date
  - Ref Date ≥ Randomization Date → Study Day = Ref Date (Randomization Date) +1

#### **Unique Subject ID**

- All subjects have unique subject ID for analyses even if a subject was enrolled after rescreened. Tables/figures/listings will be produced based on unique subject ID.
- For a rescreened subject, the unique subject ID will be derived from the first-assigned subject number though he or she seems to have multiple subject numbers in eCRF records by screening assessment. The other subject numbers, which are to be recorded within a supplemental domain, will be associated with the unique subject ID.

#### **Rescreening Subjects**

- For rescreened subjects, data collected in screening-pass visit will be used for analysis. They may have multiple records at Screening and/or Day 1 visit, which associates with a screening-pass visit and screening failure visit(s)
- Regarding a listing of SAEs in screening period, all pre-therapy SAEs captured in eCRF will be provided including screen failure records of rescreened subjects.

#### **Study Treatment Start Date**

First randomized treatment start date

#### **Study Treatment Stop Date**

- Latest end date of treatment
- Note that the end date of treatment will be captured as the end date when subjects were intended to end the treatment, rather than when subjects have actually ended the treatment.

#### Time Definitions (per GSK standard principles)

- 1 week = 7 days
- 1 month = 30.4375 days
- 1 year = 365.25 days

#### 10.6.2. Study Population

#### **Subject Disposition and Study Population**

- Screening status and reason for screening failure for a subject who has multiple subject numbers will be unique in the unique subject ID.
  - The screening status of a subject who failed screening but passed rescreening will be 'enrolled', and the reason for failure will not be counted.
  - The screening status of a subject who failed more than one screening and never passed will be 'failed', and the reason for failure will be derived from the latest failure record.
- Study population of subjects will be derived from the above unique screening status.

#### **Demographics and Baseline Characteristics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed
  as follows:
  - A date and month will be imputed as '30th June' as it will not be captured.
- Randomization date will be used as reference date of calculation.
  - o If randomization date is missing, screening date will be used.

#### Body Mass Index (BMI)

• Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

#### **Exposure**

#### **Prescribed Dose and Actual Dose**

- Prescribed dose will be derived from a dose record captured in eCRF.
- In principle, actual dose will be the same as prescribed dose except for a case in which inconsistency between a prescribed dose and prescribed bottle(s) occurs. If such an inconsistency case (e.g. wrong treatment) is detected by study team, the actual dose may be replaced with a plausible value by case-by-case review.

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
   Duration of Exposure in Days = Sum of [Exposure Duration at Each Visit]
   where Exposure Duration at Each Visit = Treatment Stop date Treatment Start date + 1
   If dose is interrupted in a visit according to dose adjustment algorithm, duration in the period will be included in duration of exposure.
- Cumulative dose will be based on the formula using prescribed dose:
   Cumulative Dose = Sum of (Exposure Duration x Dose) at Each Visit
- Daily Dose

Cumulative Dose / Duration of Exposure in Days

#### **Treatment Compliance**

Listing will include treatment compliance up to Week 4 and overall.
 Overall Compliance(%) = [(Total # of tablets actual taken)/(Total # of tablets planned

#### **Exposure**

taken)]\*100

Compliance (%) up to Week 4 = [(# of tablets actual taken up to Week 4)/(# of tablets planned taken up to Week 4)]\*100

where

Total # of tablets actual taken = Sum of (Numbers of Tablets Taken at Each Visit)

Total # of tablets planned taken = Sum of [(Treatment Stop Date – Treatment Start Date + 1) x Planned # of tablet/day in the Visit]

# of tablets actual taken up to Week 4 = Numbers of Tablets Taken of Day 1 record # of tablets planned taken up to Week 4= (Treatment Stop date of Day 1 record – Treatment Start Date of Day 1 record + 1)

Planned # of tablet/day is defined as follows according to the protocol:

- $\circ$  0 mg  $\rightarrow$  0 tablet/day
- 1 mg  $\rightarrow$  1 tablet/day
- $\circ$  2 mg  $\rightarrow$  1 tablet/day
- $\circ$  4 mg  $\rightarrow$  1 tablet/day
- $\circ$  6 mg  $\rightarrow$  1 tablet/day
- $\circ$  8 mg  $\rightarrow$  2 tablets/day
- 12 mg  $\rightarrow$  2 tablets/day
- $\circ$  18 mg  $\rightarrow$  3 tablets/day
- $\circ$  24 mg  $\rightarrow$  4 tablets/day

where dose records are derived from prescribed doses.

#### 10.6.3. Efficacy

#### **Hgb Values for Efficacy Analyses**

#### Central laboratory and HemoCue Hgb Values

For reporting purposes, central laboratory Hgb values will be used, unless otherwise specified.
 However, if a central laboratory Hgb value is missing, a corresponding non-missing HemoCue
 Hgb value, which is associated with the identical subject number and visit, will be used.

#### **Evaluable Hgb Values**

- Note that this will not be applicable for reporting summaries and figures, but applicable for reporting listings.
- Evaluable Hgb values will be based on on-therapy central laboratory and/or HemoCue Hgb values that are not taken within the 8 weeks following a transfusion or within the 8 weeks following a non-randomized ESA medication (except protocol-specified ESA treatment in screening period).

If an Hgb record meets at least one following criteria, the Hgb record will have a flag of evaluable Hgb = 'N'.

 ○ Blood Product Administration Date < Date of Hgb data ≤ Blood Product Administration Date + 56 (days)

#### **Hgb Values for Efficacy Analyses**

ESA Start Date < Date of Hgb data ≤ ESA Stop Date + 56 (days)</li>

#### Flowchart for Hgb efficacy analyses



 Basically, scheduled visits between Day 1 and Week 24 will be applicable to this flowchart, but analyses including by-visit summaries may include other schedued visits (ie. screening and follow-up visit).

[1] Regarding partially evaluated Hgb values, the following summaries of Hgb will include a unscheduled visit:

- Summary of Number (%) of subjects who have an Hgb level of less than 7.5 g/dL
- Summary of Number (%) of subjects who have an Hgb level of more than 13.0 g/dL and number of episodes

#### Hgb increase of more than 2 g/dL over any 4 weeks

- For this reporting purpose, Hgb values from central laboratory will be used as previously described.
- A subject who has at least one record with Hgb increase of more than 2 g/dL over any 4 weeks will be counted.
- Hgb increase will be calculated for scheduled visits between Day 1 and Week 24 if available (i.e. Week 4 Hgb Day 1 Hgb, Week 8 Hgb Week 4 Hgb, ...)

Illustration of calculation (example in case of Week 12 missing)

| Hgb<br>(g/dL) | Lab Date | Study<br>Day | Visit | Hgb increase |
|---------------|-----------|--------------|---------|----------------|
| 9.1 | 01FEB2017 | 1 | Day 1 | Not calculated |
| 9.8 | 02MAR2017 | 30 | Week 4 | 0.7 |
| 11.9 | 02APR2017 | 61 | Week 8 | 2.1 |
| 12.6 | 07JUN2017 | 127 | Week 16 | Not calculated |
| 12.7 | 08JUL2017 | 158 | Week 20 | 0.1 |
| 12.3 | 02AUG2017 | 183 | Week 24 | -0.4 |

#### Scatter plot of Hgb assessments: Central Laboratory vs. HemoCue

 All available pairs of Hgb (i.e. non-missing values in both from central laboratory and from the corresponding HemoCue measurement) will be used. The figure will include Pearson's

#### **Hgb Values for Efficacy Analyses**

correlation coefficient.

#### Scatter plot of Change from Baseline in Hgb at Week 4 vs. Candidate Covariates

- The following scatter plot figures will be produced for overall and dialysis status groups:
  - Change from baseline in Hgb at Week 4 vs. Body Weight at Screening
  - Change from baseline in Hgb at Week 4 vs. Baseline Hgb
- Vertical axis will indicate the change from baseline in Hgb (g/dL) at Week 4, horizontal axis will
  indicate the candidate covariates; body weight (kg) at screening or baseline Hgb (g/dL).

#### Scatter plot of Mean Dose during Week 12 to 24 vs. Candidate Covariates

- The following scatter plot figures will be produced for overall and dialysis status groups:
  - Mean Dose during Week 12 to 24 vs. Body Weight at Screening
  - Mean Dose during Week 12 to 24 vs. Baseline Hgb
- Vertical axis will indicate the mean dose (mg), horizontal axis will indicate the candidate covariates; body weight (kg) at screening or baseline Hgb (g/dL).
- Mean dose will be calculated from the arithmetic mean using the latest 3 exposure records (i.e., for completers Week 12, 16, and 20), which are based on the prescribed doses and the scheduled visits.
- Subjects who has less than 3 dosing records will be excluded from the figures.
- Mean dose during Week 12 to 24 will also be summarized and listed.

#### **Dose Adjustment**

#### Dose adjustment algorithm

- Dose Adjustment algorithm will be based on HemoCue Hgb values at scheduled visits. No Hgb values measured at unscheduled visits will be included.
- Dose will be derived from prescribed dose recorded in eCRF, not actual dose associated with container numbers.
- The following table illustrates the algorithm using analysis flags as below:
  - (FL\_A): Adjustment flags will be counted if prescribed dose recorded in eCRF is changed from that of the previous visit.
  - o (FL\_B): Over 13 g/dL flags will be counted if HemoCue Hgb >13 g/dL is observed.
  - o (FL C): Interruption flags will be counted if prescribed dose recorded in eCRF is zero.

Treatment durations will be calculated based on the following formula:

Duration (days) = Treatment Stop Date – Treatment Start Date + 1

#### Illustration of dose adjustment algorithm

| | Treatment | | HemoCue | | (FL_A) | (FL_B) | (FL_C) |
|---|---|---|---|---|---|---|---|
| Visit | Start date/ | | Hgb | Dose | Adjust- | Over | Inter- |
| (Example) | Stop date | Duration | (g/dL) | (mg) | ment | 13 g/dL | ruption |
| Day 1 | 01FEB2017/ | 29 | 11.1 | 4 | N | N | N |
| | 01MAR2017 | | | | | | |
| Week 4 | 02MAR2017/ | 14 | 11.4 | 4 | N | N | N |

| Dose A | Adjustment | | | | | | | |
|--------|------------|-------------------------|----|------|---|---|---|---|
| | | 15MAR2017 | | | | | | |
| | Week 8 | 02APR2017/<br>01MAY2017 | 30 | 11.8 | 2 | Υ | N | N |
| | Week 12 | 02MAY2017/<br>01JUN2017 | 31 | 13.4 | 0 | Y | Υ | Y |
| | Week 16 | 02JUN2017/<br>01JUL2017 | 30 | 11.6 | 1 | Y | N | N |
| | Week 20 | 02JUL2017/<br>01AUG2017 | 31 | 12.7 | 0 | Υ | N | Υ |
| | Week 24 | - | - | 12.3 | - | - | N | - |

For summary tables, how to use flags is described within the next items;

- 'Duration (days) of treatment interruption due to Hgb >13 g/dL'
- > 'Dose adjustment'

#### Duration (days) of treatment interruption due to Hgb >13 g/dL

Calculation of duration of treatment interruption due to Hgb >13 g/dL will be based on the above algorithm and the below formula.

Duration (days) = Sum of [Duration]<sub>n</sub>

where

[Duration]<sub>n</sub> represents exposure duration at visit n.

If over 13 g/dL flag (FL\_B) = 'Y' and interruption flag (FL\_C) = 'Y':

Duration (days) = Treatment Stop Date - Treatment Start Date + 1

If else:

Duration (days) = 0

#### Frequency of dose adjustment

Calculation of frequency of dose adjustment will be based on the above algorithm.

- Number of dose adjustment will be counted for each subject as follows:
  - Counts of adjustment flag = 'Y'

#### Number of dose adjustment to reach the lower Hgb target (10.0 g/dL)

Number of dose adjustment to reach the lower Hgb target will be counted for each subject as follows

• Counts of adjustment flag ='Y' at visits before Date to reach the lower Hgb target, including a record which firstly achieved the lower Hgb target.

#### **Iron Endpoints**

#### Subjects who used i.v. and oraliron

- Number of subjects who used i.v. and/or oral iron will be summarized
- Subjects who used i.v. and oral iron will be defined as follows:
  - Subjects with on-therapy i.v. and/or oral iron medication collected in a specific eCRF form (CONMEDS-IRON).

#### **Quarterly IV Iron Dose**

- Records of on-therapy iron medication will be used for the following calculations
- Monthly average i.v. iron by quarter = Total i.v. iron dose during each quarter (mg) / (duration in a quarter (days) / 30.4375 days).
- Total i.v. iron dose during each quarter (mg) will be carried with the following formula using each record. Duration will be derived from iron medication start/stop date:
  - Total i.v. iron dose in each quarter (mg) = (iron dose<sub>1</sub>\*frequency<sub>1</sub>\*duration<sub>1</sub>) + ... + (iron dose<sub>n</sub>\*frequency<sub>n</sub>\*duration<sub>n</sub>)
  - $\circ$  Duration (days) = (stop date<sub>1</sub> start date<sub>1</sub> + 1) + ... + (stop date<sub>n</sub> start date<sub>n</sub> + 1) Frequency is defined as follows:
    - If subject receives iron dose with once daily → frequency = 1
    - o If subject receives iron dose with BID → frequency = 2
    - o If subject receives iron dose with TID → frequency = 3
    - o If subject receives iron dose with QID → frequency = 4
- Quarters will be defined as follows:
  - Quarter 1:start date = Randomization Date
     end date = Treatment Start Date at Week 12 1 (day)
  - Quarter 2:start date = Treatment Start Date at Week 12
     end date = Study Treatment Stop Date
  - If treatment start date at Week 12 is missing (i.e. early withdrawal before Week 12), the end date of Quarter 1 will be replaced with Study Treatment Stop Date.
     Quarter 2 will not be generated.
  - Iron medication start/stop date will be defined newly for the analyses in addition to Quarter start/end date to derive amount of iron dose within a specified quarter (analysis flags may be used to judge which quarters the iron records should belong to).
- If iron medication start date < randomization date, the iron medication start date will be replaced with randomization date for the analyses.
- If iron medication end date > Study Treatment Stop Date, the iron medication stop date will be replaced with Study Treatment Stop Date for the analyses.
  - If iron medication start date and stop date step over quarters, the iron medication record will be divided; the end date in the former record and the start date in the latter record will be replaced with the quarter end date and the next quarter start date, respectively.

| Quarter State of Iron Medication | Definition |
|---|---|
| Quarter 1 | Iron Medication End Date ≤ Quarter 1 End Date |
| Quarter 2 | Quarter 2 Start Date ≤ Iron Medication Start Date |
| Quarter 1 & 2 (will be divided as described above) | Iron Medication Start Date ≤ Quarter 1 End Date and |
| | Quarter 2 Start Date ≤ Iron Medication Stop Date |

#### NOTES:

- Only on-therapy iron medication will be evaluated.
- If no start or stop date is recorded on iron medication, the date will be replaced with Randomization Date or Study Treatment Stop Date, respectively.

#### **TIBC**

- TIBC will be calculated automatically by the central laboratory using:
  - TIBC = UIBC + total iron

#### **TSAT**

- Based on literature review the distribution of TSAT is skewed and requires a log-transformation. Calculation of statistics on log-transformed data are described in Section 10.5.2.2.
- TSAT will be calculated automatically by the central laboratory using:
  - O TSAT = 100 \* (Serum Iron/TIBC)

#### Hepcidin

 Based on literature review the distribution of hepcidin is skewed and requires a logtransformation. Calculation of statistics on log-transformed data are described in Section 10.5.2.2.

#### 10.6.4. Safety

#### **Adverse Events**

#### AE up to Week 4

Cut-off date of Week 4 for individuals will be based on Week 4 visit date which is associated with the earliest date throughout Week 4 records (i.e., SDTM.SVSTDTC).

#### **AE of Special Interest**

AEs of special interest are manually-selected at patient-level (i.e. following case-by-case review by members of the SRT including representatives from the local Japan team) and not at preferred term level.

Adverse events of special interest are classified as follows:

- Thrombosis and/or tissue ischemia secondary to excessive erythropoiesis
- Death, MI, stroke, heart failure, thromboembolic events, thrombosis of vascular access
- Cardiomyopathy
- Pulmonary artery hypertension
- Cancer-related mortality and tumor progression and recurrence
- Esophageal and gastric erosions
- Proliferative retinopathy, macular edema, choroidal neovascularization
- Exacerbation of rheumatoid arthritis

#### **CV** Events

Basically, patient profiles of CV events will be provided according to records captured in eCRF, except for Peripheral Arterial Thrombosis Embolism (PAT) form.

CV events in PAT form will be provided only when a related AE sequence number is not present. This is because several records in PAT form are captured just for AESI information, instead of CV events.

#### **Laboratory Parameters**

#### **Imputation**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - $\circ$  Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - $\circ$  Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - $\circ$  Example 3: 0 Significant Digits = '< x' becomes x 1
- The following laboratory values will not be applicable for this imputation:
  - o Hgb, serum iron, serum ferritin, serum transferrin, TIBC, UIBC, TSAT, and Hepcidin
- The default convention for reporting of clinical laboratory units will be the international system of units (SI units).

#### Log-transformation

Lipid parameters will be log-transformed and the percent change from baseline will be reported.
 Based on literature review the distributions of hepcidin and TSAT are skewed and require a log-transformation. Other endpoints may also be log-transformed if deemed appropriate (See Section 10.5.2.2).

#### **Others**

Just for summaries of PCI cutoffs, the absolute neutrophils and lymphocytes count will be calculated by multiplying the percentages given for each subject by the absolute white blood count.

#### 10.6.5. Pharmacokinetic

#### Dose level

- Summaries by dose level and used tablet strength will be based on an actual dose associated with a container number. (See Section 10.6.2). Tablet strength is defined as follows:
  - Actual dose =  $0 \text{ mg} \rightarrow 0 \text{ mg}$  tablet strength
  - Actual dose = 1 mg  $\rightarrow$  1 mg tablet strength
  - Actual dose =  $2 \text{ mg} \rightarrow 2 \text{ mg}$  tablet strength
  - Actual dose =  $4 \text{ mg} \rightarrow 4 \text{ mg}$  tablet strength

- Actual dose = 6 mg  $\rightarrow$  6 mg tablet strength
- Actual dose =  $8 \text{ mg} \rightarrow 4 \text{ mg}$  tablet strength
- Actual dose = 12 mg → 6 mg tablet strength
- O Actual dose = 18 mg → 6 mg tablet strength
- O Actual dose = 24 mg → 6 mg tablet strength
- Dose level will be derived from an actual dose of the visit (including unscheduled visits) which meets the following:
  - Treatment Start Date ≤ Date of last dose taken prior to PK sampling ≤ Treatment Stop Date

#### **Others**

- Dose normalized PK parameters will be derived from [PK parameters/actual dose (mg)].
- In pooled analyses, data collected in Week 12 and Week 24 will be aggregated.
- For the PK parameters calculation, the concentration at 0 hr and 7 hr will be set to 0.
- Individual's PK parameters calculated less than 4 time point concentration or any time deviated (beyond  $\pm$  30 min of scheduled timepoints) concentration will be omitted from summaries and figures.

## 10.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

#### 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as completing all periods of the study including the follow-up visit. |
| | The study will be completed with the last subject's last study visit |
| | Withdrawn subjects will not be replaced in the study. |
| | All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |

### 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

#### 10.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Concomitant<br>Medications<br>/Dialysis | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

#### 10.7.2.2. Handling of Missing Data for Statistical Analysis

If a central laboratory Hgb value is missing, a corresponding non-missing HemoCue Hgb value will be used. Any other imputation will not be conducted for Hgb.

## 10.8. Appendix 8: Values of Potential Clinical Importance

## 10.8.1. Laboratory Values

| Laboratory Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Low Flag | High Flag |
| Albumin (serum) | g/L | < 30 g/L | >55 g/L |
| Aspartate Aminotransferase | IU/L | N/A | ≥ 3x ULRR |
| Alanine Aminotransferase | IU/L | N/A | ≥ 3x ULRR |
| Bilirubin (total) | μmol/L | N/A | ≥ 2x ULRR |
| Calcium (albumin-adjusted) | mmol/L | < 1.87 mmol/L | > 2.56 mmolL |
| Bicarbonate (total) | mmol/L | < 20 mmol/L | > 32 mmol/L |
| Inorganic phosphate | mmol/L | < 0.81 mmol/L | > 1.77 mmol/L |
| Potassium (serum) | mmol/L | < 0.5 mmol/L below<br>LLRR | > 1.0 mmol/L above<br>ULRR |
| Sodium (serum) | mmol/L | < 130 mmol/L | > 150 mmol/L |

| Laboratory Parameter | Units | Clinical Concern Range | |
|----------------------|-------|------------------------|----------------|
| | | Low Flag (< x) | High Flag (>x) |
| Platelet Count | GI/L | < 80 GI/L | > 500 GI/L |
| WBC Count | GI/L | < 1x LLRR | >5x ULRR |
| Neutrophils | GI/L | < 1.0 GI/L | N/A |
| Lymphocytes | GI/L | < 0.5 GI/L | N/A |

| Laboratory Parameter | Units | Clinical Concern Range | |
|----------------------|-------|------------------------|----------------|
| | | Low Flag (< x) | High Flag (>x) |
| Ferritin | μg/L | < 100 μg/L | > 1200 μg/L |
| TSAT | % | <15 % | >40 % |
| iPTH | ng/L | N/A | > 9x ULRR |

## 10.8.2. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 mmHg | > 180 mmHg |
| Diastolic Blood Pressure | mmHg | < 45 mmHg | > 110 mmHg |
| Heart Rate | beats/min | < 40 beats/min | > 110 beats/min |

## 10.9. Appendix 9: Multicenter Studies

It is anticipated that subject accrual will be spread thinly across centers and summaries of data by center would be unlikely to be informative. Therefore, data from all participating centers will be just pooled prior to analysis.

## 10.10. Appendix 10: Examination of Covariates, Subgroups & Other Strata

#### 10.10.1. Handling of Covariates, Subgroups & Other Strata

- The following is a list of covariates that may be used in descriptive summaries by subgroups.
- Additional covariates of clinical interest may also be considered.
- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be refined prior to database freezing.

| Category | Covariates and / or Subgroups |
|---|---|
| Covariates <sup>[1]</sup> | Body Weight (kg) at Screening |
| | Baseline Hgb (g/dL) |
| Subgroup | Dialysis Status |
| | <ul> <li>Newly started dialysis (Dialysis newly started &lt; 12 weeks<br/>before screening): Patients not using ESAs after the start<br/>of dialysis</li> </ul> |
| | Maintenance dialysis (Dialysis started >= 12 weeks before screening): Patients not using ESAs within 8 weeks before screening (including interruption of ESA therapy) |

<sup>[1]</sup> This category will be used only to produce exploratory figures of scatter plot.

## 10.11. Appendix 11: Multiple Comparisons & Multiplicity

## 10.11.1. Handling of Multiple Comparisons & Multiplicity

There is no hypothesis to be tested.

# 10.12. Appendix 12: Model Checking and Diagnostics for Statistical Analyses

There is no statistical analysis assumption.

## 10.13. Appendix 13 – Abbreviations & Trade Marks

## 10.13.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| $CV_b/CV_w$ | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| Hgb | Hemoglobin |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| IP | Investigational Product |
| IV | Intravenous |
| GUI | Guidance |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| TIBC | Total Iron Binding Capacity |
| TSAT | Transferrin Saturation |
| UIBC | Unsaturated Iron Binding Capacity |
| GSK | GlaxoSmithKline |

#### 10.13.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies | Trademarks not owned by the GlaxoSmithKline Group of Companies |
|---|---|
| N/A | WinNonlin |
| | SAS |
| | HemoCue |

## 10.14. Appendix 14: List of Data Displays

#### 10.14.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|------------------------|-------------|
| Study Population | 1.1 to 1.32 | N/A |
| Efficacy | 2.1 to 2.48 | 2.1 to 2.16 |
| Safety | 3.1 to 3.46 | 3.1 |
| Pharmacokinetic | 4.1 to 4.8 4.1 to 4.15 | |
| Section | Listings | |
| ICH Listings | 1 to 28 | |
| Other Listings | 29 t | o 69 |

#### 10.14.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in 10.15: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

## 10.14.3. Study Population Tables

| Study | Population Ta | ables | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | SAC |
| Subjec | t Disposition | | | | |
| 1.1. | Assigned | ES8 | Summary of Subject Status and Reason for Study Withdrawal | ICH E3, GSK CTR, FDAAA, EudraCT | Y |
| 1.2. | Assigned | ES8 | Summary of Subject Status and Reason for Study Withdrawal by Dialysis Status | | Υ |
| 1.3. | All Treated<br>Subjects | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | Y |
| 1.4. | All<br>Screening | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | Υ |
| 1.5. | Enrolled | NS1 | Summary of Subjects Enrolled by Country and Site ID | EudraCT/clinical operations | Υ |
| Protoc | ol Deviations | | | | |
| 1.6. | Assigned | DV1 | Summary of Important Protocol Deviations | ICH E3 | Υ |
| 1.7. | Assigned | IE1 | Summary of Inclusion/Exclusion Criteria Deviations | ICH E3 | Υ |
| Popula | ations Analys | ed | | | |
| 1.8. | All<br>Screening | SP1 | Summary of Study Populations | IDSL | Y |
| 1.9. | Assigned | SP2A | Summary of Exclusions from All Treated Subjects Population | IDSL | Υ |
| Demog | Demographic and Baseline Characteristics | | | | |
| 1.10. | All Treated<br>Subjects | DM1 | Summary of Demographic Characteristics | ICH E3, GSK CTR, FDAAA, EudraCT | Y |
| 1.11. | All Treated<br>Subjects | DM1 | Summary of Demographic Characteristics by Dialysis Status | | Y |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | SAC |
| 1.12. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | Υ |
| 1.13. | All Treated<br>Subjects | DM5 | Summary of Race and Racial Combinations | ICH E3, GSK CTR, FDAAA, EudraCT | Y |
| 1.14. | All Treated<br>Subjects | FH1 | Summary of Family History for CV Risk Factors | IDSL | Υ |
| 1.15. | All Treated<br>Subjects | SU1 | Summary of Substance Use (History of Tobacco Use, Alcohol Intake) | IDSL | Y |
| Prior a | nd Concomit | ant Medications | | | |
| 1.16. | All Treated<br>Subjects | MH4 | Summary of Current Medical Conditions | ICH E3 | Υ |
| 1.17. | All Treated<br>Subjects | MH4 | Summary of Current Medical Conditions by Dialysis Status | | Υ |
| 1.18. | All Treated<br>Subjects | MH4 | Summary of Past Medical Conditions | ICH E3 | Y |
| 1.19. | All Treated<br>Subjects | MH4 | Summary of Past Medical Conditions by Dialysis Status | | Y |
| 1.20. | All Treated<br>Subjects | CM1 | Summary of Concomitant Medications (Prior-Treatment) | ICH E3 | Y |
| 1.21. | All Treated<br>Subjects | CM1 | Summary of Concomitant Medications (On-therapy) | ICH E3 | Y |
| 1.22. | All Treated<br>Subjects | CM1 | Summary of Concomitant Medications (Post-therapy) | ICH E3 | Y |
| 1.23. | All Treated<br>Subjects | CM1 | Summary of Other Concomitant Medication (On-therapy) | | Y |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | SAC |
| 1.24. | All Treated<br>Subjects | CM1 | Summary of Other Concomitant Medication by Dialysis Status (Ontherapy) | | Y |
| 1.25. | All Treated<br>Subjects | POP_T1 | Summary of Blood Products and Blood Supportive Care Products (Ontherapy) | | Υ |
| 1.26. | All Treated<br>Subjects | POP_T1 | Summary of Blood Products and Blood Supportive Care Products by Dialysis Status (On-therapy) | | Y |
| Dialysi | is | | | | |
| 1.27. | All Treated<br>Subjects | POP_T2 | Summary of Dialysis Status | | Y |
| 1.28. | All Treated<br>Subjects | POP_T3 | Summary of Baseline Hemodialysis | | Υ |
| 1.29. | All Treated<br>Subjects | POP_T4 | Summary of Baseline Vascular Access | | Υ |
| Expos | ure and Treat | ment Compliand | ce | | |
| 1.30. | All Treated<br>Subjects | POP_T5 | Summary of Exposure to Study Treatment | ICH E3 | Υ |
| 1.31. | All Treated<br>Subjects | POP_T5 | Summary of Exposure to Study Treatment by Dialysis Status | | Υ |
| 1.32. | All Treated<br>Subjects | POP_T6 | Summary of Treatment Compliance | | Υ |

## 10.14.4. Efficacy Tables

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | SAC |
| Hgb | | | | | |
| 2.1. | All Treated<br>Subjects | EFF_T1 | Summary of Change from Baseline in Hgb by Visit | | Υ |
| 2.2. | All Treated<br>Subjects | EFF_T1 | Summary of Change from Baseline in Hgb by Visit by Dialysis Status | | Υ |
| 2.3. | All Treated<br>Subjects | EFF_T2 | Summary of Number (%) of subjects by Hgb change from baseline category at Week 4 | | Υ |
| 2.4. | All Treated<br>Subjects | EFF_T2 | Summary of Number (%) of subjects by Hgb change from baseline category at Week 4 by Dialysis Status | | Υ |
| 2.5. | All Treated<br>Subjects | EFF_T1 | Summary of Hgb by Visit | | Υ |
| 2.6. | All Treated<br>Subjects | EFF_T1 | Summary of Hgb by Visit by Dialysis Status | | Υ |
| 2.7. | All Treated<br>Subjects | EFF_T3 | Summary of Number (%) of subjects with Hgb within the target range by Visit | | Υ |
| 2.8. | All Treated<br>Subjects | EFF_T3 | Summary of Number (%) of subjects with Hgb within the target range by Visit by Dialysis Status | | Υ |
| 2.9. | All Treated<br>Subjects | EFF_T4 | Summary of Time (in days) to reach the lower target Hgb level (10.0 g/dL) | | Υ |
| 2.10. | All Treated<br>Subjects | EFF_T4 | Summary of Time (in days) to reach the lower target Hgb level (10.0 g/dL) by Dialysis Status | | Υ |
| 2.11. | All Treated<br>Subjects | EFF_T5 | Summary of Number (%) of subjects who have an Hgb level of less than 7.5 g/dL | | Υ |
| Efficac | Efficacy: Tables | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | SAC | | | |
| 2.12. | All Treated<br>Subjects | EFF_T5 | Summary of Number (%) of subjects who have an Hgb level of less than 7.5 g/dL by Dialysis Status | | Υ | | | |
| 2.13. | All Treated<br>Subjects | EFF_T5 | Summary of Number (%) of subjects who have an Hgb increase of more than 2.0 g/dL over any 4 weeks | | Υ | | | |
| 2.14. | All Treated<br>Subjects | EFF_T5 | Summary of Number (%) of subjects who have an Hgb increase of more than 2.0 g/dL over any 4 weeks | | Y | | | |
| 2.15. | All Treated<br>Subjects | EFF_T6 | Summary of Number (%) of subjects who have an Hgb level of more than 13.0 g/dL and number of episodes by Dialysis Status | | Υ | | | |
| 2.16. | All Treated<br>Subjects | EFF_T6 | Summary of Number (%) of subjects who have an Hgb level of more than 13.0 g/dL and number of episodes by Dialysis Status | | Y | | | |
| Iron Us | se | | | | | | | |
| 2.17. | All Treated<br>Subjects | EFF_T7 | Summary of Dose of i.v. iron during the treatment period | | Y | | | |
| 2.18. | All Treated<br>Subjects | EFF_T7 | Summary of Dose of i.v. iron during the treatment period by Dialysis Status | | Υ | | | |
| 2.19. | All Treated<br>Subjects | EFF_T8 | Summary of Number (%) of subjects who use iron during the treatment period | | Υ | | | |
| 2.20. | All Treated<br>Subjects | EFF_T8 | Summary of Number (%) of subjects who use iron during the treatment period by Dialysis Status | | Y | | | |
| Iron Pa | arameters (fer | ritin, TSAT, hep | cidin, serum iron, and TIBC) | | | | | |
| 2.21. | All Treated<br>Subjects | LB1 | Summary of Ferritin (ug/L) by Visit | Includes Baseline values | Y | | | |
| 2.22. | All Treated<br>Subjects | LB1 | Summary of Ferritin (ug/L) by Visit by Dialysis Status | Includes Baseline values | Y | | | |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | SAC |
| 2.23. | All Treated<br>Subjects | LB1 | Summary of Ferritin (ug/L) Change from Baseline by Visit | | Υ |
| 2.24. | All Treated<br>Subjects | LB1 | Summary of Ferritin (ug/L) Change from Baseline by Visit by Dialysis Status | | Y |
| 2.25. | All Treated<br>Subjects | EFF_T9 | Summary of Transferrin Saturation (%) by Visit | Includes Baseline values | Y |
| 2.26. | All Treated<br>Subjects | EFF_T9 | Summary of Transferrin Saturation (%) by Visit by Dialysis Status | Includes Baseline values | Y |
| 2.27. | All Treated<br>Subjects | EFF_T10 | Summary of Transferrin Saturation (%) Percent Change from Baseline by Visit | | Y |
| 2.28. | All Treated<br>Subjects | EFF_T10 | Summary of Transferrin Saturation (%) Percent Change from Baseline by Visit by Dialysis Status | | Y |
| 2.29. | All Treated<br>Subjects | EFF_T9 | Summary of Hepcidin (nmol/L) by Visit | Includes Baseline values | Y |
| 2.30. | All Treated<br>Subjects | EFF_T9 | Summary of Hepcidin (nmol/L) by Visit by Dialysis Status | Includes Baseline values | Y |
| 2.31. | All Treated<br>Subjects | EFF_T10 | Summary of Hepcidin (nmol/L) Percent Change from Baseline by Visit | | Y |
| 2.32. | All Treated<br>Subjects | EFF_T10 | Summary of Hepcidin (nmol/L) Percent Change from Baseline by Visit by Dialysis Status | | Y |
| 2.33. | All Treated<br>Subjects | LB1 | Summary of Serum Iron (umol/L) by Visit | Includes Baseline values | Y |
| 2.34. | All Treated<br>Subjects | LB1 | Summary of Serum Iron (umol/L) by Visit by Dialysis Status | Includes Baseline values | Y |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | SAC |
| 2.35. | All Treated<br>Subjects | LB1 | Summary of Serum Iron (umol/L) Change from Baseline by Visit | | Y |
| 2.36. | All Treated<br>Subjects | LB1 | Summary of Serum Iron (umol/L) Change from Baseline by Visit by Dialysis Status | | Y |
| 2.37. | All Treated<br>Subjects | LB1 | Summary of Total Iron Binding Capacity (umol/L) by Visit | Includes Baseline values | Y |
| 2.38. | All Treated<br>Subjects | LB1 | Summary of Total Iron Binding Capacity (umol/L) by Visit by Dialysis Status | Includes Baseline values | Y |
| 2.39. | All Treated<br>Subjects | LB1 | Summary of Total Iron Binding Capacity (umol/L) Change from Baseline by Visit | | Y |
| 2.40. | All Treated<br>Subjects | LB1 | Summary of Total Iron Binding Capacity (umol/L) Change from Baseline by Visit by Dialysis Status | | Y |
| Dose a | djustment | | | | |
| 2.41. | All Treated<br>Subjects | EFF_T11 | Summary of Dose level (mg) by Visit | Includes mean dose (mg) during Week 12 to 24 | Y |
| 2.42. | All Treated<br>Subjects | EFF_T11 | Summary of Dose level (mg) by Visit by Dialysis Status | Includes mean dose (mg) during Week 12 to 24 | Y |
| 2.43. | All Treated<br>Subjects | EFF_T12 | Summary of Duration (days) of treatment interruption due to Hgb >13.0 g/dL | | Y |
| 2.44. | All Treated<br>Subjects | EFF_T12 | Summary of Duration (days) of treatment interruption due to Hgb >13.0 g/dL by Dialysis Status | | Y |
| 2.45. | All Treated<br>Subjects | EFF_T13 | Summary of Dose Adjustment | | Y |
| 2.46. | All Treated | EFF_T13 | Summary of Dose Adjustment by Dialysis Status | | Y |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | SAC |
| | Subjects | | | | |
| 2.47. | All Treated<br>Subjects | EFF_T14 | Summary of Number (%) of Subjects with Each Dose Level by Visit | | Y |
| 2.48. | All Treated<br>Subjects | EFF_T14 | Summary of Number (%) of Subjects with Each Dose Level by Visit by Dialysis Status | | Y |

# 10.14.5. Efficacy Figures

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | SAC |
| Hgb | | | | | |
| 2.1. | All Treated<br>Subjects | EFF_F1 | Plot of Mean Hgb (g/dL) and 95% CI for Change from Baseline over Time | | Υ |
| 2.2. | All Treated<br>Subjects | EFF_F1 | Plot of Mean Hgb (g/dL) and 95% CI for Change from Baseline over Time by Dialysis Status | | Y |
| 2.3. | All Treated<br>Subjects | EFF_F1 | Plot of Mean Hgb (g/dL) and 95% CI over Time | | Υ |
| 2.4. | All Treated<br>Subjects | EFF_F1 | Plot of Mean Hgb (g/dL) and 95% CI over Time by Dialysis Status | | Υ |
| 2.5. | All Treated<br>Subjects | EFF_F2 | Figure of Number (%) of subjects with Hgb within the target range over time | Like Fig. 2.7.6.2.3.1-2 in NESP CTD 2.7.6 | Υ |
| 2.6. | All Treated<br>Subjects | EFF_F2 | Figure of Number (%) of subjects with Hgb within the target range over time by Dialysis Status | | Υ |
| 2.7. | All Treated<br>Subjects | EFF_F3 | Kaplan-Meier plot of Time (in days) to reach the lower target Hgb level (10.0 g/dL) | | Υ |
| 2.8. | All Treated<br>Subjects | EFF_F3 | Kaplan-Meier plot of Time (in days) to reach the lower target Hgb level (10.0 g/dL) by Dialysis Status | | Υ |
| 2.9. | All Treated<br>Subjects | EFF_F4 | Scatter plot of Hgb assessments: Central Laboratory vs. HemoCue | | Y |
| Dose A | Adjustment | | | | |
| 2.10. | All Treated<br>Subjects | EFF_F5 | Histogram of GSK1278863 Dose by Visit | | Y |

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | SAC |
| 2.11. | All Treated<br>Subjects | EFF_F6 | Subject Profiles of Hgb and Dose over Time | | Υ |
| Iron Pa | arameters | | | | |
| 2.12. | All Treated<br>Subjects | EFF_F1 | Plot of Mean and 95% CI for Ferritin Change from Baseline over time | | Y |
| 2.13. | All Treated<br>Subjects | EFF_F1 | Plot of Geometric Mean and 95% CI for Transferrin Saturation Percent Change from Baseline over time | | Y |
| 2.14. | All Treated<br>Subjects | EFF_F1 | Plot of Geometric Mean and 95% CI for Hepcidin Percent Change from Baseline over time | | Y |
| 2.15. | All Treated<br>Subjects | EFF_F1 | Plot of Mean and 95% CI for Serum Iron Change from Baseline over time | | Y |
| 2.16. | All Treated<br>Subjects | EFF_F1 | Plot of Mean and 95% CI for Total Iron Binding Capacity Change from Baseline over time | | Y |
| Other | | | | | |
| 2.17. | All Treated<br>Subjects | EFF_F7 | Scatter Plot of Change from Baseline in Hgb at Week 4 vs. Body Weight | | Y |
| 2.18. | All Treated<br>Subjects | EFF_F7 | Scatter Plot of Change from Baseline in Hgb at Week 4 vs. Body Weight by Dialysis Status | | Y |
| 2.19. | All Treated<br>Subjects | EFF_F7 | Scatter Plot of Change from Baseline in Hgb at Week 4 vs. Baseline Hgb | | Y |
| 2.20. | All Treated<br>Subjects | EFF_F7 | Scatter Plot of Change from Baseline in Hgb at Week 4 vs. Baseline Hgb by Dialysis Status | | Y |
| 2.21. | All Treated<br>Subjects | EFF_F7 | Scatter Plot of Mean Dose during Week 12 to 24 vs. Body Weight | | Y |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | SAC |
| 2.22. | All Treated<br>Subjects | EFF_F7 | Scatter Plot of Mean Dose during Week 12 to 24 vs. Body Weight by Dialysis Status | | Y |
| 2.23. | All Treated<br>Subjects | EFF_F7 | Scatter Plot of Mean Dose during Week 12 to 24 vs. Baseline Hgb | | Y |
| 2.24. | All Treated<br>Subjects | EFF_F7 | Scatter Plot of Mean Dose during Week 12 to 24 vs. Baseline Hgb by Dialysis Status | | Y |

# 10.14.6. Safety Tables

| Safety | afety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | SAC |
| Advers | Adverse Events (AEs) | | | | |
| 3.1. | All Treated<br>Subjects | AE1 | Summary of On-Therapy AEs by SOC and PT | ICH E3 | Y |
| 3.2. | All Treated<br>Subjects | AE1 | Summary of On-Therapy AEs by SOC and PT by Dialysis Status | | Y |
| 3.3. | All Treated<br>Subjects | AE5 | Summary of On-Therapy AEs by SOC and PT and Maximum Intensity | ICH E3 | Y |
| 3.4. | All Treated<br>Subjects | AE1 | Summary of On-Therapy AEs up to Week 4 by SOC and PT | ICH E3 | Y |
| 3.5. | All Treated<br>Subjects | AE1 | Summary of On-Therapy AEs up to Week 4 by SOC and PT by Dialysis Status | | Y |
| 3.6. | All Treated<br>Subjects | AE5 | Summary of On-Therapy AEs up to Week 4 by SOC and PT and Maximum Intensity | ICH E3 | Y |
| 3.7. | All Treated<br>Subjects | AE1 | Summary of Post-Therapy AEs by SOC and PT | ICH E3 | Y |
| 3.8. | All Treated<br>Subjects | AE5 | Summary of Post-Therapy AEs by SOC and PT and Maximum Intensity | ICH E3 | Y |
| 3.9. | All Treated<br>Subjects | AE1 | Summary of On-Therapy Drug-Related AEs by SOC and PT | ICH E3 | Y |
| 3.10. | All Treated<br>Subjects | AE1 | Summary of On-Therapy Drug-Related AEs by SOC and PT by Dialysis Status | | Y |
| 3.11. | All Treated<br>Subjects | AE5 | Summary of On-Therapy Drug-Related AEs by SOC and PT and Maximum Intensity | ICH E3 | Υ |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | SAC |
| 3.12. | All Treated<br>Subjects | AE1 | Summary of On-Therapy Drug-Related AEs up to Week 4 by SOC and PT | ICH E3 | Υ |
| 3.13. | All Treated<br>Subjects | AE1 | Summary of On-Therapy Drug-Related AEs up to Week 4 by SOC and PT by Dialysis Status | | Υ |
| 3.14. | All Treated<br>Subjects | AE5 | Summary of On-Therapy Drug-Related AEs up to Week 4 by SOC and PT and Maximum Intensity | ICH E3 | Y |
| 3.15. | All Treated<br>Subjects | AE1 | Summary of Post-Therapy Drug-Related AEs by SOC and PT | ICH E3 | Υ |
| 3.16. | All Treated<br>Subjects | AE5 | Summary of Post-Therapy Drug-Related AEs by SOC and PT and Maximum Intensity | ICH E3 | Υ |
| 3.17. | All Treated<br>Subjects | AE15 | Summary of On-Therapy Common (>=5%) Non-Serious AEs by SOC and PT (Subjects & No. of Occurrences) | FDAAA, EudraCT | Y |
| Seriou | s and Other S | ignificant AEs | | | |
| 3.18. | All Treated<br>Subjects | AE1 | Summary of On-Therapy Serious AEs | GSK CTR | Υ |
| 3.19. | All Treated<br>Subjects | AE1 | Summary of Post-Therapy Serious AEs | GSK CTR | Υ |
| 3.20. | All Treated<br>Subjects | AE16 | Summary of Serious AEs by SOC and PT (Subjects & No. of Occurrences) | FDAAA, EudraCT | Υ |
| 3.21. | All Treated<br>Subjects | AE1 | Summary of AEs Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment by SOC and PT | IDSL | Υ |
| AEs of | Special Inter | est | | | |
| 3.22. | All Treated<br>Subjects | SAFE_T1 | Summary of On-Therapy AEs of special interest | | Y |
| 3.23. | All Treated | SAFE_T1 | Summary of On-Therapy AEs of special interest by Dialysis Status | | Υ |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | SAC |
| | Subjects | | | | |
| 3.24. | All Treated<br>Subjects | SAFE_T1 | Summary of Post-Therapy AEs of special interest | | Υ |
| Labora | tory Chemist | ry | | | |
| 3.25. | All Treated<br>Subjects | LB1 | Summary of Chemistry Values by Visit | ICH E3<br>Includes Baseline values | Υ |
| 3.26. | All Treated<br>Subjects | LB1 | Summary of Chemistry Changes from Baseline by Visit | ICH E3 | Υ |
| 3.27. | All Treated<br>Subjects | SAFE_T2 | Summary of Percent change from Baseline in Lipid Parameters (total cholesterol, LDL cholesterol and HDL cholesterol) by Visit | | Υ |
| 3.28. | All Treated<br>Subjects | LB15 | Summary of Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | Υ |
| 3.29. | All Treated<br>Subjects | LB17 | Summary of Worst Case Chemistry Results Relative to PCI Criteria Post-Baseline Relative to Baseline | ICH E3 | Y |
| Hemate | ology | | | | |
| 3.30. | All Treated<br>Subjects | LB1 | Summary of Hematology Values by Visit | ICH E3<br>Includes Baseline values | Y |
| 3.31. | All Treated<br>Subjects | LB1 | Summary of Hematology Changes from Baseline by Visit | ICH E3 | Y |
| 3.32. | All Treated<br>Subjects | LB15 | Summary of Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | Y |
| 3.33. | All Treated<br>Subjects | LB17 | Summary of Worst Case Hematology Results Relative to PCI Criteria Post-Baseline Relative to Baseline | ICH E3 | Y |
| Other I | _aboratory Te | ests | | | |
| 3.34. | All Treated | LB1 | Summary of Other Laboratory Values by Visit | ICH E3 | Y |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | SAC |
| | Subjects | | | Includes Baseline values | |
| 3.35. | All Treated<br>Subjects | LB1 | Summary of Other Laboratory Changes from Baseline by Visit | ICH E3 | Y |
| 3.36. | All Treated<br>Subjects | LB15 | Summary of Worst Case Other Laboratory Results Relative to Normal Range Post-Baseline Relative to Baselinet | ICH E3 | Y |
| 3.37. | All Treated<br>Subjects | LB17 | Summary of Worst Case Other Laboratory Results Relative to PCI Criteria Post-Baseline Relative to Baseline | ICH E3 | Y |
| Hepato | biliary (Liver) | 1 | | | |
| 3.38. | All Treated<br>Subjects | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | IDSL | Y |
| 3.39. | All Treated<br>Subjects | LIVER10 | Summary of Subjects Meeting Emergent Hepatobiliary Laboratory Abnormality Criteria | IDSL<br>Listing may be sufficient if few events. | Y |
| ECG | | | | | |
| 3.40. | All Treated<br>Subjects | EG1 | Summary of ECG Findings | IDSL | Y |
| 3.41. | All Treated<br>Subjects | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | Y |
| Vital Si | gns | | | | |
| 3.42. | All Treated<br>Subjects | SAFE_T3<br>based on VS1 | Summary of Vital Signs by Visit | Summarized by each assessment status (i.e. pre-dialysis and post-dialysis) | Y |
| 3.43. | All Treated<br>Subjects | SAFE_T3<br>based on VS1 | Summary Change from Baseline in Vital Signs by Visit | Summarized by each assessment status (i.e. pre-dialysis and post-dialysis) | Y |
| 3.44. | All Treated<br>Subjects | SAFE_T4<br>based on VS7 | Summary of Worst Case Vital Sign Results Relative to PCI Criteria Post-Baseline Relative to Baseline | Summarized by each assessment status (i.e. pre-dialysis and post-dialysis) | Y |
| Ophtha | almology | | | | |

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | SAC |
| 3.45. | All Treated<br>Subjects | SAFE_T5 | Summary of Ophthalmologic Exams at Screening | | Υ |
| 3.46. | All Treated<br>Subjects | SAFE_T6 | Summary of On-Therapy Ophthalmologic Exams | | Υ |
| Safety | Summaries for | or a Plain Languaç | ge Summary | | |
| 3.47. | All Treated<br>Subjects | AE3 | Summary of On-Therapy Serious Drug-Related AEs | | Υ |
| 3.48. | All Treated<br>Subjects | AE3 | Summary of On-Therapy Non-Serious Drug-Related AEs | | Y |

## 10.14.7. Safety Figures

| Safety | Safety : Figures | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | SAC |
| Clinica | l Laboratory | Analyses | | | |
| 3.1. | All Treated<br>Subjects | SAFE_F1 | Plot of Percent change from Baseline in Lipid Parameters (total cholesterol, LDL cholesterol, and HDL cholesterol) over time | | Υ |

### 10.14.8. Pharmacokinetic Tables

| Pharmacokinetic : Tables | | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | SAC |
| Plasm | a GSK127886 | 3 Concentrations | | | |
| 4.1. | PK | PK01 | Summary of GSK1278863 Plasma Concentration by Dose level (non-transformed) | | Υ |
| 4.2. | PK | PK_T1<br>based on PK05 | Summary of GSK1278863 Plasma Concentration by Dose level (loge-transformed) | | Υ |
| PK pa | rameters | | | | |
| 4.3. | PK | PK03 | Summary of GSK1278863 Pharmacokinetic Parameters by Dose level (non-transformed) | | Υ |
| 4.4. | PK | PK05 | Summary of GSK1278863 Pharmacokinetic Parameters by Dose level (loge-transformed) | | Υ |
| 4.5. | PK | PK03 | Summary of Dose Normalized GSK1278863 Pharmacokinetic Parameters by Dose level (non-transformed) | | Υ |
| 4.6. | PK | PK05 | Summary of Dose Normalized GSK1278863 Pharmacokinetic Parameters by Dose level (loge-transformed) | | Υ |
| 4.7. | PK | PK03 | Summary of Dose Normalized GSK1278863 Pharmacokinetic Parameters by Used Tablet Strength (non-transformed) | | Υ |
| 4.8. | PK | PK05 | Summary of Dose Normalized GSK1278863 Pharmacokinetic Parameters by Used Tablet Strength (loge-transformed) | | Υ |

# 10.14.9. Pharmacokinetic Figures

| Pharm | acokinetic : | Figures | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | SAC |
| Plasm | a GSK12788 | 63 Concentrations | | | |
| 4.1. | PK | PK24 | Individual GSK1278863 Plasma Concentration-Time Plots | (Linear and Semi-Log) (by Dose) | Y |
| 4.2. | PK | PK17 | Mean GSK1278863 Plasma Concentration-Time Plots | (Linear and Semi-Log) (by Dose) | Υ |
| 4.3. | PK | PK19 | Mean (+SD) GSK1278863 Plasma Concentration-Time Plots | (Linear and Semi-Log) (by Dose) | Υ |
| 4.4. | PK | PK20 | Median GSK1278863 Plasma Concentration-Time Plots | (Linear and Semi-Log) (by Dose) | Y |
| PK Pa | rameters | | | | |
| 4.5. | PK | PK_F1 | Individual Plot of GSK1278863 Dose level and PK Parameters (AUC (0-4), AUC (0-7), Cmax) | will provide only pooled data | Y |
| 4.6. | PK | PK_F2 | Mean (+SD) Plot of GSK1278863 Dose level and PK Parameters (AUC (0-4), AUC (0-7), Cmax) | will provide only pooled data | Y |
| 4.7. | PK | PK_F3 | Median Plot of GSK1278863 Dose level and PK Parameters (AUC (0-4), AUC (0-7), Cmax) | will provide only pooled data | Y |
| 4.8. | PK | PK_F1 | Individual Plot of GSK1278863 Dose level and Dose Normalized PK Parameters (AUC (0-4), AUC (0-7), Cmax) | will provide only pooled data | Y |
| 4.9. | PK | PK_F2 | Mean (+SD) Plot of GSK1278863 Dose level and Dose Normalized PK Parameters (AUC (0-4), AUC (0-7), Cmax) | will provide only pooled data | Y |
| 4.10. | PK | PK_F3 | Median Plot of GSK1278863 Dose level and Dose Normalized PK Parameters (AUC (0-4), AUC (0-7), Cmax) | will provide only pooled data | Y |
| 4.11. | PK | PK_F4 | Box Plot of GSK1278863 Dose level and Dose Normalized PK Parameters (AUC (0-4), AUC (0-7), Cmax) | will provide only pooled data | Y |
| 4.12. | PK | PK_F1 | Individual Plot of GSK1278863 Used Tablet Strength and Dose Normalized PK Parameters (AUC (0-4), AUC (0-7), Cmax) | will provide only pooled data | Y |

| Pharmacokinetic : Figures | | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | SAC |
| 4.13. | PK | PK_F2 | Mean (+SD) Plot of GSK1278863 Used Tablet Strength and Dose Normalized PK Parameters (AUC (0-4), AUC (0-7), Cmax) | will provide only pooled data | Υ |
| 4.14. | PK | PK_F3 | Median Plot of GSK1278863 Used Tablet Strength and Dose<br>Normalized PK Parameters (AUC (0-4), AUC (0-7), Cmax) | will provide only pooled data | Υ |
| 4.15. | PK | PK_F4 | Box Plot of GSK1278863 Used Tablet Strength and Dose<br>Normalized PK Parameters (AUC (0-4), AUC (0-7), Cmax) | will provide only pooled data | Υ |

## 10.14.10. ICH Listings

| | | | ICH : Listings | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | SAC |
| Study | Populations | | | | |
| Subjec | ct Disposition | | | | |
| 1. | Assigned | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | Υ |
| 2. | All Treated<br>Subjects | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | Υ |
| 3. | All Screening | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | Y |
| Protoc | ol Deviations | | | | |
| 4. | Assigned | DV2 | Listing of Important Protocol Deviations | ICH E3 | Υ |
| 5. | Assigned | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | Υ |
| Popula | ations Analysed | | | | |
| 6. | Assigned | SP3 | Listing of Subjects Excluded from All Treated Subjects Population | ICH E3 Note: IDSL shell for SP3a in development. e.g., subjects screened but not randomized, subjects randomized but not treated, subjects with deviations leading to exclusion from per protocol population (can be separate listing per population). | Y |
| Demog | graphic and Base | eline Charact | teristics | | |
| 7. | All Treated<br>Subjects | DM2 | Listing of Demographic Characteristics | ICH E3 | Y |
| 8. | All Treated<br>Subjects | DM9 | Listing of Race | ICH E3 | Y |

| | | | ICH : Listings | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | SAC |
| Dialysi | ialysis | | | | |
| 9. | All Treated<br>Subjects | POP_L1 | Listing of Dialysis Status | | Υ |
| Exposi | ure and Treatme | nt Compliand | ce | | |
| 10. | All Treated<br>Subjects | POP_L2<br>based on<br>EX3 | Listing of Exposure Data | ICH E3 | Υ |
| 11. | All Treated<br>Subjects | POP_L3 | Listing of Treatment Compliance | ICH E3 Up to Week 4 and overall compliance will be provided. | Υ |
| Efficac | у | | | | |
| Hgb | | | | | |
| 12. | All Treated<br>Subjects | EFF_L1 | Listing of Hgb Data | | Υ |
| 13. | All Treated<br>Subjects | EFF_L2 | Listing of Subjects who have an Hgb level of less than 7.5 g/dL | | Υ |
| 14. | All Treated<br>Subjects | EFF_L2 | Listing of Subjects who have an Hgb increase of more than 2.0 g/dL over any 4 weeks | | Υ |
| 15. | All Treated<br>Subjects | EFF_L2 | Listing of Subjects who have an Hgb increase of more than 13.0 g/dL | | Υ |
| 16. | All Treated<br>Subjects | LB5 | Listing of Iron Parameter Data | Ferritin, TSAT, hepcidin, serum iron, and TIBC will be included. | Υ |
| Safety | | | | | |

| | | | ICH : Listings | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | SAC |
| Advers | se Events | | | | |
| 17. | All Treated<br>Subjects | AE8 | Listing of All Adverse Events | ICH E3 | Y |
| 18. | All Treated<br>Subjects | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | Υ |
| 19. | All Treated<br>Subjects | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | Υ |
| Seriou | s and Other Sigr | nificant Adve | rse Events | | |
| 20. | All Treated<br>Subjects | AE8 | Listing of Fatal Serious Adverse Events | ICH E3 Fatal and Non-Fatal SAEs are combined into a single listing for ClinPharm studies (i.e., "Listing of Serious Adverse Events"). | Υ |
| 21. | All Treated<br>Subjects | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3 Fatal and Non-Fatal SAEs are combined into a single listing for ClinPharm studies (i.e., "Listing of Serious Adverse Events"). | Y |
| 22. | All Screening | AE8 | Listing of Serious AEs in Screening Period | All pre-therapy SAEs captured in eCRF will be provided including screen failure records of rescreened subjects. | Y |
| 23. | All Treated<br>Subjects | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | Y |
| 24. | All Treated<br>Subjects | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | Υ |

| | | | ICH : Listings | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | SAC |
| 25. | All Treated<br>Subjects | SAFE_L1 | Listing of Adverse Events of Special Interest | ICH E3 Displays will be produced with AESI category in addition of AE8 template. | Υ |
| All Lab | oratory | | | | |
| 26. | All Treated<br>Subjects | LB5 | Listing of All Chemistry Data for Subjects with Any Value Outside of Normal Range/of PCI | ICH E3 May be split into separate listings by chemistry, hematology, urinalysis, etc. Display ALL labs for a subject who experienced a value of potential clinical concern/importance. | Y |
| 27. | All Treated<br>Subjects | LB5 | Listing of All Hematology Data for Subjects with Any Value Outside of Normal Range/of PCI | ICH E3 | Υ |
| 28. | All Treated<br>Subjects | LB5 | Listing of All Other Laboratory Data for Subjects with Any Value Outside of Normal Range/of PCI | ICH E3 | Υ |
| 29. | All Treated<br>Subjects | LB14 | Listing of Laboratory Data with Character Results | IDSL Rationale: This listing is required to ensure character laboratory results are presented. | Υ |

# 10.14.11. Non-ICH Listings

| Non-IC | Non-ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | SAC |
| Study | Study Population | | | | |
| Demog | graphic and Bas | seline Characteri | istics | | |
| 30. | All Treated<br>Subjects | FH4 | Listing of Family Members with History of Cardiovascular Risk Factors | | Υ |
| 31. | All Treated<br>Subjects | SU2 | Listing of Substance Use History | | Υ |
| Prior a | nd Concomitar | nt Medications | | | |
| 32. | All Treated<br>Subjects | MH2 | Listing of Medical Conditions | | Y |
| 33. | All Treated<br>Subjects | CM2 | Listing of Concomitant Medications | | Y |
| 34. | All Treated<br>Subjects | POP_L4 | Listing of ESA Concomitant Medications | | Y |
| 35. | All Treated<br>Subjects | POP_L5 | Listing of Iron Concomitant Medications | | Y |
| 36. | All Treated<br>Subjects | POP_L6 | Listing of Blood Products and Blood Supportive Care Products | | Y |
| Dialys | is | | | | |
| 37. | All Treated<br>Subjects | POP_L7 | Listing of Baseline Hemodialysis and Changes in Hemodialysis | | Y |
| 38. | All Treated<br>Subjects | POP_L8 | Listing of Baseline Vascular Access | | Y |

| Non-IC | SH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | SAC |
| 39. | All Treated<br>Subjects | POP_L9 | Listing of Subjects with Vascular Therapeutic Procedures during the Study Period | | Υ |
| Efficac | ;y | | | | |
| Safety | | | | | |
| Suicida | ality-Related Ad | dverse Event | | | |
| 40. | All Treated<br>Subjects | IDSL standard | Listing of Possible Suicidality-Related Adverse Event Data: Event and Description (Sections 1-2) | | Y |
| 41. | All Treated<br>Subjects | IDSL standard | Listing of Possible Suicidality-Related Adverse Event Data: Possible Cause(s) (Section 3) | | Υ |
| 42. | All Treated<br>Subjects | IDSL standard | Listing of Possible Suicidality-Related Adverse Event Data: (Section 4) | | Υ |
| 43. | All Treated<br>Subjects | IDSL standard | Listing of Possible Suicidality-Related Adverse Event Data: (Section 5-8) | | Υ |
| Clinica | I Laboratory, E | CG, Vital Sign, a | nd Ophthalmology Exam | | |
| 44. | All Treated<br>Subjects | LB5 | Listing of Chemistry Data | | Υ |
| 45. | All Treated<br>Subjects | LB5 | Listing of Hematology Data | | Y |
| 46. | All Treated<br>Subjects | LB5 | Listing of Other Laboratory Data | | Y |
| 47. | All Treated<br>Subjects | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events | This listing is required for medical review of subjects with liver stopping events. | Y |
| 48. | All Treated<br>Subjects | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | This listing is required for medical review of subjects with liver stopping events. | Y |

| Non-IC | Non-ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | SAC |
| 49. | All Treated<br>Subjects | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | | Υ |
| 50. | All Treated<br>Subjects | LIVER6 | Listing of Liver Stopping Event Information for RUCAM Score | | Υ |
| 51. | All Treated<br>Subjects | LIVER7 | Listing of Liver Biopsy Details | | Υ |
| 52. | All Treated<br>Subjects | LIVER8 | Listing of Liver Imaging Details | | Υ |
| 53. | All Treated<br>Subjects | EG3 | Listing of ECG Values | | Y |
| 54. | All Treated<br>Subjects | EG5 | Listing of ECG Findings | | Υ |
| 55. | All Treated<br>Subjects | VS4 | Listing of Vital Signs | | Υ |
| 56. | All Treated<br>Subjects | VS4 | Listing of All Vital Signs for Subjects with Values of PCI | | Y |
| 57. | All Treated<br>Subjects | SAFE_L2 | Listing of Ophthalmologic Exams | | Υ |
| Pharm | Pharmacokinetic Parameters | | | | |
| 58. | PK | PK07 | Listing of GSK1278863 Pharmacokinetic Concentration-Time Data by Dose level | | Υ |
| 59. | PK | PK13 | Listing of Derived GSK1278863 Pharmacokinetic Parameters by Dose level | | Y |

## 10.14.12. Patient Profile Listings

| | | | <u>Patient Profile</u> Listings | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | SAC |
| Safety | | | | | |
| 60. | All Treated<br>Subjects | IDSL<br>standard | Patient Profile Listing of Arrhythmias | | Υ |
| 61. | All Treated<br>Subjects | IDSL<br>standard | Patient Profile Listing of Congestive Heart Failure | | Υ |
| 62. | All Treated<br>Subjects | IDSL<br>standard | Patient Profile Listing of Cerebrovascular Events/Stroke/ Transient Ischemic Attack | | Υ |
| 63. | All Treated<br>Subjects | IDSL<br>standard | Patient Profile Listing of Deep venous Thrombosis/ Pulmonary Embolism | | Υ |
| 64. | All Treated<br>Subjects | IDSL<br>standard | Patient Profile Listing of Myocardial Infarction /Unstable Angina | | Υ |
| 65. | All Treated<br>Subjects | IDSL<br>standard | Patient Profile Listing of Peripheral Arterial Thrombosis Embolism | Events will be provided only when a related AE sequence number is present (Section 10.6.4). | Υ |
| 66. | All Treated<br>Subjects | IDSL<br>standard | Patient Profile Listing of Pulmonary Hypertension | | Υ |
| 67. | All Treated<br>Subjects | IDSL<br>standard | Patient Profile Listing of Revascularization | | Y |
| 68. | All Treated<br>Subjects | IDSL<br>standard | Patient Profile Listing of Valvulopathy | | Υ |
| 69. | All Treated<br>Subjects | IDSL<br>standard | Patient Profile Listing of Deaths | | Υ |

## 10.15. Appendix 15: Example Mock Shells for Data Displays

These are provided with separated documents.

# 10.16. Appendix 16: RAP Amendment(s)

Minor wording changes are not included in below.

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 2.1 Changes to the Protocol Defined Statistical Analysis Plan | Deleted the table and added statement of "Modified text to align with the latest version of protocol as follow: 1. No interim analysis is planned. 2. The change in Hgb at Week 4 will be classified into different categories (i.e., ≤-2, >-2 to -1, >-1 to 0, >0 to 1, >1 to 2, and >2 g/dL) | Protocol was amended. 1. The interim analysis was just aiming to meet the clinical result disclosure obligation. Given our POLICY update, the due date of disclosure was changed to 'within 12 months of PCA' from 'within 8 months of PCA'. Therefore, a final analysis of 204716 study can meet the current disclosure due date. 2. Specifying the categories and ensuring there is no overlap. |
| 4 Analysis populations | The term of 'randomized population' has been changed to 'assigned population' | 'Assigned' would be more appropriate for this single arm study. |
| <ul><li>6.1.1 Planned Summary</li><li>Display Details</li><li>10.6.2 Study Population</li></ul> | Clarifications were made for a subject who has multiple numbers as follows: A subject who has multiple subject numbers (i.e. rescreened subject) will be analyzed as a unique subject based on the latest screening result. Screening status and reason for screening failure for a subject who has multiple subject numbers will be unique in the unique subject ID. Minor wording changes were also made. | Clarification |
| 7.1 Primary Efficacy<br>Analyses | Updates were made to the summaries for adding categories; within ±1 g/dL and over ±2 g/dL. | These categories would facilitate review the drug efficacy results. |
| 8 Secondary statistical analyses 10.6.3 Efficacy | It has been clarified that, on-therapy Hgb will be used for several Hgb endpoints and evaluable Hgb. In addition, 95%CI has been added to descriptive summary statistics for continuous data. | Correction and Clarification |

| Reporting and Analysis Plan_204716_Amendment_Final_V1.1 [11-Oct-2017] | | |
|---|---|---|
| Section # and Name | Description of Change | Brief Rationale |
| 8.1.2 Planned Efficacy Table Displays | Added the following clarifications in a model specification of Kaplan Meier Method: Subjects within target range at baseline will be excluded from the summary. Subjects who could not reach lower target will be regarded as censored at EoT. In addition, in dose adjustment summary, it has been clarified that what subjects will be included in summaries of duration of treatment interruption and number of dose adjustments. | Clarification |
| 8.1.2 Planned Efficacy Table Displays | Added summary tables and planed displays detail for number (%) of subjects with each dose level by visit | Tables corresponding to histogram of dose level by visit (Fig. 2.10) are necessary. |
| 8.2.1.1 Planed AE Analyses<br>Displays | <ol> <li>Clarifications were made for the maximum intensity of AEs category and how to treat different intensities in the same AE.</li> <li>It has been modified how to display serious adverse event, for both primary system organ class and preferred term.</li> </ol> | Clarification SOC for SAE summary provides a consistent presentation style that facilitates review |
| 8.2.2 Overview of Planned<br>Clinical Laboratory Analyses<br>8.2.3 Overview of Planned<br>Other Safety Analyses | Updates were made to the summaries for normal range/PCI criteria. Only the worst case results relative to normal range/PCI criteria post-baseline relative to baseline will be provided. | IDSL templates based on GSK Core<br>RAP requirements in the RAP<br>template are updated. |
| 8.2.3.1 Planned Other Safety Analyses Displays 10.5.2 Baseline Definition & Derivations 10.14.6 Safety Tables | Updates were made to the indicated sections of RAP to describe how to summarize vital sign assessment. Pre- and post-dialysis assessment will be summarized separately and non-dialysis assessment will not be summarized. | Vital sign assessment in non-dialysis day would be unlikely, so summarization would not be necessary. |
| 8.2.3.1 Planned Other Safety<br>Analyses Displays | Text added to make sure the summary display for ECG findings. | Clarification |
| 8.2.3.1 Planned Other Safety Analyses Displays | Additional summary added to ophthalmology exam, displayed along with a summary of ontherapy ophthalmology exam. No additional table is required for this update. | Worthwhile to add another way of summarization |
| 8.3.3.1 Deriving Pharmacokinetic Parameters | Modifications were made for the definition of C(last), last quantifiable concentration. | To make sure that the definitions of the parameters are consistent |
| 10.3.1 Definitions of Analysis Time Point 10.6.1 General | Text added to make sure data derivation for multiple measurements at Screening and Day 1 visit. The screening-pass visit record will be used for analysis if multiple records are present. | Clarification |

| Reporting and Analysis Plan_204716_Amendment_Final_V1.1 [11-Oct-2017] | | |
|---|---|---|
| Section # and Name | Description of Change | Brief Rationale |
| 10.4.1.3 Treatment States for<br>Concomitant Medications Data<br>10.5.3 Reporting Process &<br>Standards | Updates were made considering the case of EoT missing Further clarification has been made about descriptive summary statistics. | To ensure the definition of treatment state to cover all possible cases Clarification |
| 10.6.2 Study Population | Age Reference date for age calculation was updated Exposure Text deleted | Age Using randomization date as reference may be more appropriate rather than using screening date based on SDTM standard derivations (Note that IG suggests to only expect AGE for treated subjects, but the study expect AGE for randomized subjects). Exposure Deleted because it may not be suitable for this section |
| 10.6.3 Efficacy | Iron Endpoints: Quarterly IV Iron Dose Quarterly IV iron dose will be calculated using randomization date and EoT to support on-therapy iron definition. | To ensure that on-therapy iron and the quarterly iron are consistently defined. |
| 10.6.4 Safety | Adverse Events Corrections were made to the categories of adverse events of special interest. In a second bullet of the categories, heart failure was added and venous thromboembolism was corrected to thromboembolic events CV Events Updates were added to clarify how to provided patient profiles in PAT form. | For AEs. protocol was amended for AESI terminology. For CV events, to make sure how to output CV records based on team discussion |
| 10.6.5 Pharmacokinetic | <ol> <li>Derivation of tablet strength was clarified.</li> <li>Derivation of dose level was updated to see whether PK sampling date is included within a period of exposure for each visit as follows: <ul> <li>Treatment Start Date ≤ Date of last dose taken prior to PK sampling ≤ Treatment Stop Date</li> </ul> </li> </ol> | Clarification To make sure that the derivation can apply to an irregular PK sampling such as sampling at unscheduled visit within |

| Reporting and Analysis Plan_204716_Amendment_Final_V1.1 [11-Oct-2017] | | |
|---|---|---|
| Section # and Name | Description of Change | Brief Rationale |
| | Dose level is derived from actual dose of a visit which meets the above exposure record. | allowance of visit window. |
| 10.8 Appendix 8: Values of Potential Clinical Importance | PCI values were updated in Section 10.8.1. | To maintain consistency between global and Japan Ph3 program, use the same PCI cut off values. |
| 10.14 Appendix 14: List of Data Displays | The following bullets were modified: General Changed from 'Randomized population' to 'Assigned population' Table 1.9, Listing 6 Corrected title from 'Exclusions from Randomized Population' to 'Exclusions from All Treated Subjects Population' Table 2.13, 2.14, 2.19, 2.20, 2.43 to 2.46, 3.27, Figure 3.1 Corrected titles Table 2.47, 2.48 Added summary tables for number (%) of subjects with each dose level by visit Table 3.18, 3.19 Corrected example shell ID Table 3.42, 3.43, 3.44 Excluded statement to non-dialysis in Programming Notes of Vital Signs Listing 2,3, 22 Corrected analysis population Listing 16 Added iron parameter listing Listing 25 Deleted duplicate (listing 39) and updated IDSL example Listing 38, 39 Modified titles Listing 65 Added programming notes | Corrections and Clarifications |

| Reporting and Analysis Plan_204716_Amendment_Final_V1.2 [29-NOV-2017] | | |
|---|---|---|
| Section # and Name | Description of Change | Brief Rationale |
| 6.1 Overview of Planned Analyses | Modification was made for the title; from 'Baseline Dialysis' to 'Baseline Mode of Dialysis' | Correction |
| 8.1 Secondary Efficacy<br>Analyses | <ol> <li>Added summaries of number of dose adjustment to reach the lower Hgb target Hgb level (10.0 g/dL)</li> <li>For the summary of time to reach the lower target Hgb level, modification was made to include all subjects in the analysis.</li> </ol> | This will facilitate review of the study results Correction according to team discussion |
| 8.1.2 Planned Efficacy Table Displays | <ol> <li>Text added to clarify that the analysis of scatter plot includes Pearson's correlation coefficient.</li> <li>Updates were made to the summaries of dose level (mg) for adding P25 and P75.</li> <li>In dose adjustment summary, it has been re-corrected that all subjects including those with no dose adjustment will include a summary.</li> </ol> | <ol> <li>Clarification</li> <li>These will facilitate review of the<br/>study results.</li> <li>Reconsideration clinically for the<br/>dose adjustment summary.</li> </ol> |
| 8.2 Safety Analyses 10.14 Appendix 14: List of Data Displays | Added additional tables: On-therapy Serious Drug-Related AEs On-therapy Non-Serious Drug-Related AEs | Required for a Plain Language<br>Summary (PLS) for GSK |
| 10.4.1 Treatment States | Clarification has been made for treatment states of follow-up visit assessments. | Clarification |
| 10.6.1 General | Updates were made for definitions of treatment states; use study treatment stop date instead of end of treatment date (EoT). In addition to general changes of the treatment states due to this, note that this change has impact on the following endpoints for specific derivations: Time (in days) to reach the lower target Hgb level (10.0 g/dL) Dose of i.v. iron during the treatment period | For daprodustat, the treatment states will be more explainable on the basis of study treatment stop date derived from the exposure record rather on the basis of EoT derived from the assessment visit. |
| 10.6.2 Study Population | Text added for treatment compliance up to Week 4. | Compliance up to Week 4 will facilitate review of the study results. |
| 10.6.3 Efficacy | Deleted text that mentioned the baseline Hgb value might include that at unscheduled visits. | Missing the Hgb value at Day 1 will never happen so that no need to mention the unscheduled visits for the baseline Hgb derivation. |
| 10.6.3 Efficacy | Added the candidate covariates (body weight at screening and baseline Hgb) to provide the | This will facilitate review of |

| Reporting and Analysis Plan_204716_Amendment_Final_V1.2 [29-NOV-2017] | | |
|---|---|---|
| Section # and Name | Description of Change | Brief Rationale |
| 10.10.1 Handling of Covariates, | following scatter plot figures: | appropriateness of starting dose or |
| Subgroups & Other Strata | Change from baseline in Hgb at Week 4 vs. candidate covariates | maintenance dose. |
| 10.14.5 Efficacy Figures | Mean dose vs. candidate covariates | |
| 10.6.4 Safety | Clarification has been made for the definition of AEs up to Week 4 | Clarification and correction |
| | 2. It has been corrected how to display the CV events in PAT form. | |
| 10.6.5 Pharmacokinetic | Clarifications were made for the derivation of dose normalized PK parameters and the definition of time deviated concentration. | Clarification |